CLINICAL TRIAL: NCT02697773
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF A DOSE TITRATION REGIMEN FOR THE SUBCUTANEOUS ADMINISTRATION OF TANEZUMAB IN SUBJECTS WITH OSTEOARTHRITIS OF THE HIP OR KNEE
Brief Title: Efficacy and Safety of a Subcutaneous Tanezumab Titration Dosing Regimen in Subjects With Moderate to Severe Osteoarthritis of the Hip or Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091056; 2013-002222-23 (EudraCT Number); OA TITRATION STUDY (Other: Alias Study Number)
Record Dates: First submitted 2016-02-11; First posted 2016-03-03 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: osteoarthritis of the knee; osteoarthritis of the hip; nerve growth factor inhibitor; tanezumab
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): placebo administered subcutaneously at day 0 and week 8
  Interventions: Other: Placebo
- Tanezumab 2.5 mg (Experimental): tanezumab 2.5 mg administered subcutaneously at day 0 and week 8
  Interventions: Biological: Tanezumab 2.5 mg
- Tanezumab 2.5mg/5mg (Experimental): tanezumab 2.5 mg administered subcutaneously at day 0 and tanezumab 5 mg administered subcutaneously at week 8
  Interventions: Biological: Tanezumab 2.5mg/5mg

INTERVENTIONS:
Other: Placebo — Patient receives one dose of placebo to match tanezumab subcutaneously on Day 1 and one dose of placebo to match tanezumab subcutaneously at Week 8.
  Arms: Placebo
Biological: Tanezumab 2.5 mg — Patient receives one dose of tanezumab 2.5 mg subcutaneously on Day 1 and one dose of tanezumab 2.5 mg subcutaneously at Week 8.
  Arms: Tanezumab 2.5 mg
Biological: Tanezumab 2.5mg/5mg — Patient receives one dose of tanezumab 2.5 mg subcutaneously on Day 1 and one dose of tanezumab 5 mg subcutaneously at Week 8.
  Other Names: Titration Arm
  Arms: Tanezumab 2.5mg/5mg

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of a titration arm of tanezumab in which treatment is started at a lower dose (2.5 mg) and increased to a higher dose (5 mg) at Week 8, compared to giving 2 doses of tanezumab 2.5 mg or 2 doses of placebo. The study also evaluates the safety of the treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Osteoarthritis of the knee or hip confirmed by X-ray
* Documented history that subject tried the following medications and had insufficient pain relief or is cannot take or tolerate them: acetaminophen, NSAIDs and either tramadol or opioids
* Meet the protocol requirements for pain at screening and pain, physical function and patient global assessment of osteoarthritis at baseline
* Willing to discontinue all pain medications except study medication and rescue medication during the course of the study and use those as directed per protocol
* Women able to have children must agree to use 2 forms of contraception during the study

Exclusion Criteria:

* Body Mass Index (BMI) greater than 39
* History of diseases other than osteoarthritis in a shoulder, hip or knee (example, rheumatoid arthritis, gout, joint infections, osteonecrosis)
* Patients with x-ray showing joint conditions such as osteonecrosis (dead bone) or certain types of fractures
* Patients who have had significant trauma or surgery to a knee, hip or shoulder within the previous year
* Planned surgical procedure during the study
* Patients who are largely or wholly incapacitated (example bedridden or confined to a wheelchair, permitting little or no self-care)
* Patients who would be unwilling or unable to undergo joint replacement surgery if one eventually became necessary
* Patients with significant conditions other than osteoarthritis that could interfere with assessment of pain in the joints (example fibromyalgia, lupus erythematosus)
* Patients with significant heart, neurological or psychiatric diseases
* Patients who had cancer other than certain skin cancers within the past 5 years
* Patients with alcohol, analgesic (pain medications) or drug abuse within the past 2 years
* Women who are pregnant, breast-feeding or intending to become pregnant or breast-feed during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (87):
- United States (68):
  - Alabama Orthopaedic Surgeons, Birmingham, Alabama
  - Cahaba Research, Inc., Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Research Institute of Arizona, LLC, Surprise, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - University of Arizona Clinical and Translational Science Research Center, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Advanced Research Center, Inc, Anaheim, California
  - Medvin Clinical Research, Covina, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - Irvine Center for Clinical Research, Irvine, California
  - Robert L Freed, M.D., F.A.C.R / Clinical Interventions Research Institute, Irvine, California
  - Providence Clinical Research, North Hollywood, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Research Foundation, San Diego, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Clinical Physiology Associates, Fort Myers, Florida
  - Eastern Research, Inc., Hialeah, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - Phoenix Clinical Research, LLC, Tamarac, Florida
  - Bioclinica Research, The Villages, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Center for Advanced Research & Education (CARE), Gainesville, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Medex Healthcare Research Inc, Chicago, Illinois
  - Chicago Clinical Research Institute, Inc., Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - George Stanley Walker, MD, New Orleans, Louisiana
  - Tristan Medical Enterprises, PC dba Regeneris Medical, North Attleboro, Massachusetts
  - Michigan Orthopaedic & Spine Surgeons, Rochester Hills, Michigan
  - Arthritis and Osteoporosis Treatment and Research Center, Flowood, Mississippi
  - Office Of Stephen H. Miller, M.D., Las Vegas, Nevada
  - Arthritis And Osteoporosis Associates, Freehold, New Jersey
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Prestige Clinical Research, Franklin, Ohio
  - AC Clinical Research, Tiffin, Ohio
  - NPC Research, Oklahoma City, Oklahoma
  - Hillcrest Clinical Research, Oklahoma City, Oklahoma
  - University Orthopedics Center, State College, Pennsylvania
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Quality Medical Research, Nashville, Tennessee
  - KRK Medical Research, Arlington, Texas
  - Tekton Research, Inc, Austin, Texas
  - Urgent Care MD's, Baytown, Texas
  - Arthritis Care and Diagnostic Center, Dallas, Texas
  - T&R Clinic, PA, Fort Worth, Texas
  - Centex Studies, Inc., Houston, Texas
  - BI Research Center, Houston, Texas
  - The Pain Relief Center, Plano, Texas
  - Center for Arthritis and Rheumatic Diseases, Chesapeake, Virginia
  - Spectrum Medical, Inc, Danville, Virginia
  - National Clinical Research - Richmond, Inc, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (17):
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Manna Research Inc. (Burlington south), Burlington, Ontario
  - Dawson Road Medical Centre, Guelph, Ontario
  - Adachi Medicine Professional Corporation, Hamilton, Ontario
  - K-W Musculoskeletal Research Inc., Kitchener, Ontario
  - Western Center for Public Health and Family Medicine, London, Ontario
  - Malton Medical Centre, Mississauga, Ontario
  - Rebecca Medical Associates, Oakville, Ontario
  - King Street Medical Clinic, Oshawa, Ontario
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Diex Recheche Montreal, Inc., Montreal, Quebec
  - Recherche Clinique Sigma inc, Québec, Quebec
  - Diex Recherche Quebec Inc., Québec, Quebec
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec, Quebec
  - Centre de recherche Saint-Louis, Québec, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Puerto Rico (2):
  - Puerto Rico Medical Research Inc., Ponce, PR
  - Mindful Medical Research, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Schnitzer TJ, Conaghan PG, Berenbaum F, Abraham L, Cappelleri JC, Bushmakin AG, Viktrup L, Yang R, Brown MT. Effect size varies based on calculation method and may affect interpretation of treatment effect: an illustration using randomised clinical trials in osteoarthritis. Adv Rheumatol. 2024 Apr 22;64(1):31. doi: 10.1186/s42358-024-00358-y. PMID 38650049
- [Derived] Guermazi A, Roemer FW, Kompel AJ, Diaz LE, Crema MD, Brown MT, Hickman A, Pixton GC, Viktrup L, Fountaine RJ, Burr A, Sherlock SP, West CR. Inter-Reader Consistency and Exclusionary Findings During Radiographic Screening for Phase 3 Trials of Tanezumab in Patients With Osteoarthritis. Osteoarthr Imaging. 2022 Sep-Dec;2(3-4):100082. doi: 10.1016/j.ostima.2022.100082. Epub 2022 Nov 15. PMID 38343426
- [Derived] Ren J, Bushmakin AG, Cislo PR, Abraham L, Cappelleri JC, Dworkin RH, Farrar JT. Meaningful within-patient change for clinical outcome assessments: model-based approach versus cumulative distribution functions. J Biopharm Stat. 2025 Aug;35(5):826-838. doi: 10.1080/10543406.2023.2281575. Epub 2023 Nov 20. PMID 37982583
- [Derived] Carrino JA, McAlindon TE, Schnitzer TJ, Guermazi A, Hochberg MC, Conaghan PG, Brown MT, Burr A, Fountaine RJ, Pixton GC, Viktrup L, Verburg KM, West CR. Characterization of adverse joint outcomes in patients with osteoarthritis treated with subcutaneous tanezumab. Osteoarthritis Cartilage. 2023 Dec;31(12):1612-1626. doi: 10.1016/j.joca.2023.08.010. Epub 2023 Aug 29. PMID 37652258
- [Derived] Shoji S, Suzuki A, Nouri P, Cai CH, Gaitonde P, Marshall S. Prediction of relative change in free nerve growth factor following subcutaneous administration of tanezumab, a novel monoclonal antibody to nerve growth factor. CPT Pharmacometrics Syst Pharmacol. 2023 Sep;12(9):1358-1370. doi: 10.1002/psp4.13015. Epub 2023 Jul 31. PMID 37470295
- [Derived] Brown MT, Cornblath DR, Koltzenburg M, Gorson KC, Hickman A, Pixton GC, Gaitonde P, Viktrup L, West CR. Peripheral Nerve Safety of Nerve Growth Factor Inhibition by Tanezumab: Pooled Analyses of Phase III Clinical Studies in Over 5000 Patients with Osteoarthritis. Clin Drug Investig. 2023 Jul;43(7):551-563. doi: 10.1007/s40261-023-01286-3. Epub 2023 Jul 18. PMID 37460782
- [Derived] Colloca L, Dworkin RH, Farrar JT, Tive L, Yang J, Viktrup L, Dasic G, West CR, Whalen E, Brown MT, Gilbert SA, Verburg KM. Predicting Treatment Responses in Patients With Osteoarthritis: Results From Two Phase III Tanezumab Randomized Clinical Trials. Clin Pharmacol Ther. 2023 Apr;113(4):878-886. doi: 10.1002/cpt.2842. Epub 2023 Jan 31. PMID 36621827
- [Derived] Hunter DJ, Schnitzer TJ, Hall J, Semel D, Davignon I, Cappelleri JC, Bushmakin AG, Abraham L. Time to first and sustained improvement in WOMAC domains among patients with osteoarthritis receiving tanezumab. Osteoarthr Cartil Open. 2022 Jul 2;4(3):100294. doi: 10.1016/j.ocarto.2022.100294. eCollection 2022 Sep. PMID 36474952
- [Derived] Atkinson J, Edwards RA, Bonfanti G, Barroso J, Schnitzer TJ. A Two-Step, Trajectory-Focused, Analytics Approach to Attempt Prediction of Analgesic Response in Patients with Moderate-to-Severe Osteoarthritis. Adv Ther. 2023 Jan;40(1):252-264. doi: 10.1007/s12325-022-02336-6. Epub 2022 Oct 27. PMID 36301512
- [Derived] Mease P, Kuritzky L, Wright WL, Mallick-Searle T, Fountaine R, Yang R, Sadrarhami M, Faison W, Johnston E, Viktrup L. Efficacy and safety of tanezumab, NSAIDs, and placebo in patients with moderate to severe hip or knee osteoarthritis and a history of depression, anxiety, or insomnia: post-hoc analysis of phase 3 trials. Curr Med Res Opin. 2022 Nov;38(11):1909-1922. doi: 10.1080/03007995.2022.2113689. Epub 2022 Aug 28. PMID 35980115
- [Derived] Schnitzer TJ, Bonfanti G, Atkinson J, Donevan S, Viktrup L, Barroso J, Whalen E, Edwards RA. Characterizing 16-Week Responder Profiles Using Group-Based Trajectory Modeling in Over 4300 Clinical Trial Participants Receiving Pharmaceutical Treatment for Moderate to Severe Osteoarthritis. Adv Ther. 2022 Oct;39(10):4742-4756. doi: 10.1007/s12325-022-02290-3. Epub 2022 Aug 12. PMID 35960482
- [Derived] Conaghan PG, Dworkin RH, Schnitzer TJ, Berenbaum F, Bushmakin AG, Cappelleri JC, Viktrup L, Abraham L. WOMAC Meaningful Within-patient Change: Results From 3 Studies of Tanezumab in Patients With Moderate-to-severe Osteoarthritis of the Hip or Knee. J Rheumatol. 2022 Jun;49(6):615-621. doi: 10.3899/jrheum.210543. Epub 2022 Mar 1. PMID 35232805
- [Derived] Conaghan PG, Abraham L, Viktrup L, Cislo P. Impact of tanezumab on health status, non-work activities and work productivity in adults with moderate-to-severe osteoarthritis. BMC Musculoskelet Disord. 2022 Feb 1;23(1):106. doi: 10.1186/s12891-022-05029-x. PMID 35105318
- [Derived] Berenbaum F, Schnitzer T, Kivitz A, Viktrup L, Johnston E, Yang R, Whalen E, Tive L, Semel D. Gender, age, disease severity, body mass index and diabetes may not affect response to subcutaneous tanezumab in patients with osteoarthritis after 16 weeks of treatment. A subgroup analysis of placebo-controlled trials. Int J Clin Pract. 2021 Dec;75(12):e14975. doi: 10.1111/ijcp.14975. Epub 2021 Oct 21. PMID 34626502
- [Derived] Berenbaum F, Schnitzer TJ, Kivitz AJ, Viktrup L, Hickman A, Pixton G, Brown MT, Davignon I, West CR. General Safety and Tolerability of Subcutaneous Tanezumab for Osteoarthritis: A Pooled Analysis of Three Randomized, Placebo-Controlled Trials. Arthritis Care Res (Hoboken). 2022 Jun;74(6):918-928. doi: 10.1002/acr.24637. Epub 2022 Mar 25. PMID 33973384
- [Derived] Schnitzer TJ, Khan A, Bessette L, Davignon I, Brown MT, Pixton G, Prucka WR, Tive L, Viktrup L, West CR. Onset and maintenance of efficacy of subcutaneous tanezumab in patients with moderate to severe osteoarthritis of the knee or hip: A 16-week dose-titration study. Semin Arthritis Rheum. 2020 Jun;50(3):387-393. doi: 10.1016/j.semarthrit.2020.03.004. Epub 2020 Mar 19. PMID 32252976
- [Derived] Schnitzer TJ, Easton R, Pang S, Levinson DJ, Pixton G, Viktrup L, Davignon I, Brown MT, West CR, Verburg KM. Effect of Tanezumab on Joint Pain, Physical Function, and Patient Global Assessment of Osteoarthritis Among Patients With Osteoarthritis of the Hip or Knee: A Randomized Clinical Trial. JAMA. 2019 Jul 2;322(1):37-48. doi: 10.1001/jama.2019.8044. PMID 31265100
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4091056

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered subcutaneously on Day 1 (Baseline) and Week 8.
- Tanezumab 2.5 mg: Tanezumab (RN624 or PF-04383119) 2.5 mg injection administered subcutaneously on Day 1 (Baseline) and Week 8.
- Tanezumab 2.5/5 mg: Tanezumab (RN624 or PF-04383119) 2.5 mg injection administered subcutaneously on Day 1 (Baseline) and 5 mg injection administered subcutaneously on Week 8.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Started | 233 | 232 | 233
Treated | 232 | 231 | 233
Completed | 195 | 194 | 193
Not Completed | 38 | 38 | 40
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Death | 0 | 0 | 2
Not completed — Lack of Efficacy | 4 | 6 | 6
Not completed — Lost to Follow-up | 5 | 5 | 7
Not completed — Other | 15 | 11 | 10
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 10 | 13 | 13
Not completed — Randomized but not treated | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously.
Groups:
- Tanezumab 2.5mg/5mg: Tanezumab (RN624 or PF-04383119) 2.5 mg injection administered subcutaneously on Day 1 (Baseline) and Tanezumab 5 mg injection administered subcutaneously on Week 8.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5mg/5mg | Total
Number analyzed (Participants) | 232 | 231 | 233 | 696
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (9.8) | 60.9 (10.0) | 61.2 (9.0) | 60.83 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 145 | 151 | 453
  Male | 75 | 86 | 82 | 243
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 43 | 40 | 119
  Not Hispanic or Latino | 196 | 188 | 193 | 577
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 156 | 178 | 170 | 504
  Black or African American | 60 | 43 | 50 | 153
  Asian | 13 | 5 | 8 | 26
  Other | 3 | 5 | 5 | 13
  Unknown | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 16
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Week 16
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either Tanezumab or placebo).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale | -2.64 (0.23) | -3.23 (0.23) | -3.37 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — Step-down testing procedure within each of the primary endpoints was applied to maintain Type I error. Tanezumab 2.5/5 mg vs placebo was tested first and if found significant, then the testing was continued for Tanezumab 2.5 mg vs placebo. Tanezumab treatment group was declared as superior to placebo if the corresponding treatment contrast was significant over all 3 primary endpoints; p = 0.0129, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.60, 95% CI 2-sided [-1.07 to -0.13], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0023, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.73, 95% CI 2-sided [-1.20 to -0.26], Standard Error of Mean 0.24

2. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 16
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 17 individual questions scored on a NRS of 0 (minimum difficulty) to 10 (extreme difficulty), where higher scores indicated extreme difficulty/worse physical function.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale | -2.56 (0.22) | -3.22 (0.22) | -3.45 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed data sets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0065, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.66, 95% CI 2-sided [-1.14 to -0.19], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0002, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.89, 95% CI 2-sided [-1.37 to -0.42], Standard Error of Mean 0.24

3. Primary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis at Week 16
Description: PGA of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip (index joint) affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, where 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worsening of condition.
Time Frame: Baseline, Week 16
Population: The intent to treat population was defined as all randomized participants who received at least one dose of subcutaneous study medication (either Tanezumab or placebo).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale | -0.65 (0.08) | -0.87 (0.08) | -0.90 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0109, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.22, 95% CI 2-sided [-0.39 to -0.05], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0038, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.25, 95% CI 2-sided [-0.41 to -0.08], Standard Error of Mean 0.09

4. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Weeks 2, 4, 8 and 12
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on NRS of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Change at Week 2 | -2.20 (0.21) | -2.87 (0.21) | -2.89 (0.21)
  Change at Week 4 | -2.40 (0.21) | -3.28 (0.21) | -3.27 (0.21)
  Change at Week 8 | -2.61 (0.21) | -3.20 (0.21) | -3.02 (0.21)
  Change at Week 12 | -2.83 (0.23) | -3.61 (0.22) | -3.69 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0020, ANCOVA; Least Square Mean Difference = -0.66, 95% CI 2-sided [-1.08 to -0.24], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0014, ANCOVA; Least Square Mean Difference = -0.68, 95% CI 2-sided [-1.10 to -0.26], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.88, 95% CI 2-sided [-1.31 to -0.45], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.87, 95% CI 2-sided [-1.30 to -0.44], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0085, ANCOVA; Least Square Mean Difference = -0.59, 95% CI 2-sided [-1.03 to -0.15], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0657, ANCOVA; Least Square Mean Difference = -0.41, 95% CI 2-sided [-0.85 to 0.03], Standard Error of Mean 0.22
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0012, ANCOVA; Least Square Mean Difference = -0.78, 95% CI 2-sided [-1.25 to -0.31], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority; p = 0.0004, ANCOVA; Least Square Mean Difference = -0.86, 95% CI 2-sided [-1.33 to -0.38], Standard Error of Mean 0.24

5. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 24
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either Tanezumab or placebo). Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline | 7.30 (1.15) | 7.08 (1.16) | 7.33 (1.26)
  Change at Week 24: number analyzed (Participants) | 185 | 200 | 202
  Change at Week 24 | -3.07 (2.43) | -2.80 (2.50) | -2.95 (2.49)

6. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Weeks 2, 4, 8 and 12
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Change at Week 2 | -2.14 (0.21) | -2.89 (0.21) | -3.05 (0.21)
  Change at Week 4 | -2.28 (0.21) | -3.30 (0.21) | -3.38 (0.21)
  Change at Week 8 | -2.55 (0.21) | -3.17 (0.21) | -3.12 (0.21)
  Change at Week 12 | -2.75 (0.22) | -3.61 (0.22) | -3.80 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0004, ANCOVA; Least Mean Square Difference = -0.75, 95% CI 2-sided [-1.17 to -0.34], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.91, 95% CI 2-sided [-1.33 to -0.50], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.02, 95% CI 2-sided [-1.45 to -0.60], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.11, 95% CI 2-sided [-1.53 to -0.68], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0057, ANCOVA; Least Square Mean Difference = -0.63, 95% CI 2-sided [-1.07 to -0.18], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p = 0.0114, ANCOVA; Least Square Mean Difference = -0.57, 95% CI 2-sided [-1.02 to -0.13], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12:Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0004, ANCOVA; Least Square Mean Difference = -0.86, 95% CI 2-sided [-1.33 to -0.38], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.05, 95% CI 2-sided [-1.52 to -0.58], Standard Error of Mean 0.24

7. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 24
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 17 individual questions scored on a NRS of 0 (minimum difficulty) to 10 (extreme difficulty), where higher scores indicated maximum difficulty/worse physical function.
Time Frame: Baseline, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline | 7.38 (1.12) | 7.18 (1.11) | 7.39 (1.18)
  Change at Week 24: number analyzed (Participants) | 185 | 200 | 202
  Change at Week 24 | -3.03 (2.37) | -2.85 (2.51) | -3.01 (2.46)

8. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8 and 12
Description: PGA of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip (index joint) affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, where 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities).
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Change at Week 2 | -0.74 (0.07) | -0.91 (0.07) | -0.87 (0.07)
  Change at Week 4 | -0.75 (0.07) | -1.01 (0.07) | -0.97 (0.07)
  Change at Week 8 | -0.82 (0.07) | -0.97 (0.07) | -0.91 (0.07)
  Change at Week 12 | -0.83 (0.08) | -1.01 (0.08) | -1.11 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0236, ANCOVA; Least Mean Square Difference = -0.17, 95% CI 2-sided [-0.32 to -0.02], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis subscale and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0958, ANCOVA; Least Square Mean Difference = -0.12, 95% CI 2-sided [-0.27 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0007, ANCOVA; Least Square Mean Difference = -0.26, 95% CI 2-sided [-0.40 to -0.11], Standard Error of Mean 0.07
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0040, ANCOVA; Least Mean Square Difference = -0.21, 95% CI 2-sided [-0.36 to -0.07], Standard Error of Mean 0.07
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0498, ANCOVA; Least Square Mean Difference = -0.15, 95% CI 2-sided [-0.31 to -0.00], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.2380, ANCOVA; Least Square Mean Difference = -0.09, 95% CI 2-sided [-0.24 to 0.06], Standard Error of Mean 0.08
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0426, ANCOVA; Least Square Mean Difference = -0.17, 95% CI 2-sided [-0.34 to -0.01], Standard Error of Mean 0.09
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p = 0.0014, ANCOVA; Least Square Mean Difference = -0.28, 95% CI 2-sided [-0.45 to -0.11], Standard Error of Mean 0.09

9. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis at Week 24
Description: PGA of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip (index joint) affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, where 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worse condition.
Time Frame: Baseline, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline | 3.46 (0.57) | 3.42 (0.60) | 3.53 (0.62)
  Change at Week 24: number analyzed (Participants) | 185 | 200 | 202
  Change at Week 24 | -0.87 (0.85) | -0.72 (0.93) | -0.91 (1.03)

10. Secondary Outcome: Percentage of Participants Meeting Outcomes Measures in Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index
Description: Participants were considered as OMERACT-OARSI responders: if the change (improvement) from baseline to week of interest was greater than or equal to (>=) 50 percent and greater or equal to (>=) 2 units in either WOMAC pain subscale or physical function subscale score; if change (improvement) from baseline to week of interest was >=20 percent and >=1 unit in at least 2 of the following: 1) WOMAC pain subscale score, 2) WOMAC physical function subscale score, 3) PGA of osteoarthritis. WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [extreme pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [extreme difficulty], higher score = worse physical function) and PGA of osteoarthritis (score: 1 [very good] to 5 [very poor], higher score = worse condition). Missing data was imputed using mixed baseline/last observation carried forward (BOCF/LOCF).
Time Frame: Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
percentage of participants
  Week 2 | 50.4 | 65.4 | 67.4
  Week 4 | 58.6 | 74.0 | 74.7
  Week 8 | 61.6 | 67.5 | 69.5
  Week 12 | 66.4 | 77.5 | 81.1
  Week 16 | 65.1 | 72.7 | 79.0
  Week 24: number analyzed (Participants) | 185 | 200 | 202
  Week 24 | 68.1 | 66.5 | 68.8
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Odds ratio and 95% confidence interval (CI) estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0027, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.22 to 2.61]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.36 to 2.89]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Odds ratio and 95% confidence interval (CI) estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.33 to 2.95]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 10, analysis 3]; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.37 to 3.04]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Odds ratio and 95% confidence interval (CI) estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.2283, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.86 to 1.87]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.1066, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.93 to 2.03]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Odds ratio and 95% confidence interval (CI) estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0154, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.10 to 2.54]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.38 to 3.27]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Odds ratio and 95% confidence interval (CI) estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.1139, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.92 to 2.07]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 10, analysis 9]; Test type: Superiority; p = 0.0014, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.31 to 3.04]

11. Secondary Outcome: Percentage of Participants Achieving Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Reduction >= 30 Percent (%), >=50%, >=70% and >=90% Response
Description: Percentage of participants with reduction in WOMAC pain intensity of at least (>=) 30%, 50%, 70% and 90% at Weeks 2, 4, 8, 12, 16 and 24 compared to baseline were classified as responders to WOMAC pain subscale and are reported here. WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Week 2, 4, 8, 12, 16 and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
percentage of participants
  Week 2: At least 30% reduction | 38.8 | 56.3 | 56.2
  Week 2: At least 50% reduction | 22.8 | 38.5 | 38.2
  Week 2: At least 70% reduction | 15.5 | 25.5 | 24.5
  Week 2: At least 90% reduction | 6.9 | 13.4 | 9.4
  Week 4: At least 30% reduction | 47.0 | 65.4 | 63.5
  Week 4: At least 50% reduction | 30.2 | 48.5 | 48.5
  Week 4: At least 70% reduction | 16.4 | 29.4 | 29.6
  Week 4: At least 90% reduction | 8.2 | 16.0 | 15.5
  Week 8: At least 30% reduction | 49.1 | 61.9 | 61.4
  Week 8: At least 50% reduction | 30.2 | 47.2 | 42.5
  Week 8: At least 70% reduction | 17.2 | 30.3 | 25.8
  Week 8: At least 90% reduction | 9.1 | 13.0 | 12.9
  Week 12: At least 30% reduction | 54.3 | 70.1 | 75.1
  Week 12: At least 50% reduction | 40.5 | 60.2 | 56.2
  Week 12: At least 70% reduction | 24.1 | 39.8 | 39.5
  Week 12: At least 90% reduction | 9.9 | 18.6 | 18.9
  Week 16: At least 30% reduction | 54.7 | 68.0 | 70.4
  Week 16: At least 50% reduction | 37.9 | 54.5 | 57.1
  Week 16: At least 70% reduction | 25.0 | 34.6 | 36.5
  Week 16: At least 90% reduction | 9.5 | 14.7 | 14.2
  Week 24: At least 30% reduction: number analyzed (Participants) | 185 | 200 | 202
  Week 24: At least 30% reduction | 60.5 | 60.5 | 59.9
  Week 24: At least 50% reduction: number analyzed (Participants) | 185 | 200 | 202
  Week 24: At least 50% reduction | 39.5 | 40.0 | 41.6
  Week 24: At least 70% reduction: number analyzed (Participants) | 185 | 200 | 202
  Week 24: At least 70% reduction | 23.2 | 21.0 | 21.3
  Week 24: At least 90% reduction: number analyzed (Participants) | 185 | 200 | 202
  Week 24: At least 90% reduction | 10.3 | 10.5 | 8.9
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0009, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.30 to 2.78]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.36 to 2.90]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0015, Regression, Logistic; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.29 to 2.96]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.34 to 3.07]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0251, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.07 to 2.75]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0276, Regression, Logistic; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.06 to 2.72]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0404, Regression, Logistic; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.03 to 3.71]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p = 0.3486, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.70 to 2.72]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.42 to 3.02]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.32 to 2.79]
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.41 to 3.05]
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.46 to 3.15]
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0024, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.28 to 3.18]
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 13]; Test type: Superiority; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.35 to 3.34]
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0172, Regression, Logistic; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.14 to 3.72]
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 15]; Test type: Superiority; p = 0.0173, Regression, Logistic; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.14 to 3.72]
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0118, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.11 to 2.35]
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 2.5/5 mg; Week 8, >=30%:Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0132, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [1.10 to 2.32]
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.35 to 2.92]
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 2.5/5 mg; Week 8, >=50%:Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0100, Regression, Logistic; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.13 to 2.45]
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0023, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.28 to 3.12]
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 21]; Test type: Superiority; p = 0.0322, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.04 to 2.58]
Statistical Analysis 23: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.2005, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.81 to 2.67]
Statistical Analysis 24: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 23]; Test type: Superiority; p = 0.1923, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.82 to 2.68]
Statistical Analysis 25: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0013, Regression, Logistic; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.28 to 2.79]
Statistical Analysis 26: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 25]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.50, 95% CI 2-sided [1.68 to 3.73]
Statistical Analysis 27: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.45 to 3.10]
Statistical Analysis 28: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 27]; Test type: Superiority; p = 0.0014, Regression, Logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.26 to 2.67]
Statistical Analysis 29: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.33 to 2.99]
Statistical Analysis 30: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 29]; Test type: Superiority; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.37 to 3.06]
Statistical Analysis 31: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0127, Regression, Logistic; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.16 to 3.49]
Statistical Analysis 32: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 31]; Test type: Superiority; p = 0.0075, Regression, Logistic; Odds Ratio (OR) = 2.11, 95% CI 2-sided [1.22 to 3.64]
Statistical Analysis 33: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16 >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0061, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.17 to 2.52]
Statistical Analysis 34: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 33]; Test type: Superiority; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.33 to 2.88]
Statistical Analysis 35: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16 >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority — The two comparisons for 'Participants with >=50% reduction from baseline in WOMAC Pain at Week 16' (tanezumab 2.5 mg treatment group versus placebo and tanezumab 2.5/5 mg treatment group versus placebo) were adjusted for multiple comparisons using the Hochberg procedure and an overall significance level of 0.05; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.29 to 2.76]
Statistical Analysis 36: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0411, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.02 to 2.31]
Statistical Analysis 37: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 36]; Test type: Superiority; p = 0.0090, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.14 to 2.57]
Statistical Analysis 38: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.1149, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.89 to 2.86]
Statistical Analysis 39: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 38]; Test type: Superiority; p = 0.1351, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.87 to 2.79]
Statistical Analysis 40: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 11, analysis 35]; Test type: Superiority — The two comparisons for 'Participants with ≥50% reduction from baseline in WOMAC Pain at Week 16' (tanezumab 2.5 mg treatment group versus placebo and tanezumab 2.5/5 mg treatment group versus placebo) were adjusted for multiple comparisons using the Hochberg procedure and an overall significance level of 0.05; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.17, 95% CI 2-sided [1.48 to 3.16]

12. Secondary Outcome: Percentage of Participants With Cumulative Percent Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 16
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a NRS of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain. Percentage of participants with cumulative reduction (as percent) (greater than 0% ; >= 10, 20, 30, 40, 50, 60, 70, 80 and 90%; = 100 %) in WOMAC pain subscale from Baseline to Week 16 were reported, participants (%) are reported more than once in categories specified. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
percentage of participants
  >=0% | 82.3 | 87.4 | 88.4
  >=10% | 79.3 | 81.8 | 85.4
  >=20% | 65.5 | 74.0 | 79.0
  >=30% | 54.7 | 68.0 | 70.4
  >=40% | 45.7 | 63.2 | 66.1
  >=50% | 37.9 | 54.5 | 57.1
  >=60% | 31.5 | 44.2 | 44.6
  >=70% | 25.0 | 34.6 | 36.5
  >=80% | 17.2 | 24.2 | 27.0
  >=90% | 9.5 | 14.7 | 14.2
  =100% | 3.9 | 8.2 | 10.7

13. Secondary Outcome: Percentage of Participants Achieving Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Reduction >= 30 Percent (%), >=50%, >=70% and >=90% Response
Description: Percentage of participants with reduction in WOMAC physical function of at least (>=) 30%, 50%, 70% and 90% at weeks 2, 4, 8, 12, 16 and 24 compared to baseline were classified as responders to WOMAC physical function subscale. WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. Physical function refers to participant's ability to move around and perform usual activities of daily living. WOMAC physical function subscale: 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint (knee or hip) during past 48 hours,calculated as mean of the scores from 17 individual questions scored on a NRS of 0 (minimum difficulty) to 10 (extreme difficulty), where higher scores indicated extreme difficulty/worse physical function. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
percentage of participants
  Week 2: At least 30% reduction | 35.8 | 55.8 | 56.7
  Week 2: At least 50% reduction | 23.7 | 35.1 | 39.9
  Week 2: At least 70% reduction | 12.1 | 26.4 | 24.9
  Week 2: At least 90% reduction | 5.2 | 11.3 | 9.0
  Week 4: At least 30% reduction | 45.7 | 66.7 | 64.4
  Week 4: At least 50% reduction | 26.7 | 48.1 | 48.5
  Week 4: At least 70% reduction | 15.1 | 30.3 | 30.5
  Week 4: At least 90% reduction | 6.9 | 13.4 | 14.6
  Week 8: At least 30% reduction | 47.8 | 58.9 | 61.8
  Week 8: At least 50% reduction | 28.9 | 47.6 | 42.5
  Week 8: At least 70% reduction | 16.8 | 27.3 | 27.9
  Week 8: At least 90% reduction | 7.8 | 13.0 | 12.9
  Week 12: At least 30% reduction | 53.0 | 70.1 | 75.1
  Week 12: At least 50% reduction | 37.9 | 57.1 | 56.2
  Week 12: At least 70% reduction | 22.0 | 38.5 | 39.5
  Week 12: At least 90% reduction | 9.1 | 17.7 | 18.0
  Week 16: At least 30% reduction | 54.3 | 65.8 | 71.7
  Week 16: At least 50% reduction | 36.6 | 54.1 | 57.1
  Week 16: At least 70% reduction | 22.8 | 34.2 | 36.1
  Week 16: At least 90% reduction | 10.3 | 14.3 | 14.6
  Week 24: At least 30% reduction: number analyzed (Participants) | 185 | 200 | 202
  Week 24: At least 30% reduction | 57.3 | 58.0 | 58.4
  Week 24: At least 50% reduction: number analyzed (Participants) | 185 | 200 | 202
  Week 24: At least 50% reduction | 38.4 | 36.5 | 41.6
  Week 24: At least 70% reduction: number analyzed (Participants) | 185 | 200 | 202
  Week 24: At least 70% reduction | 21.1 | 22.0 | 20.8
  Week 24: At least 90% reduction: number analyzed (Participants) | 185 | 200 | 202
  Week 24: At least 90% reduction | 8.1 | 10.5 | 8.4
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.45 to 3.11]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.32, 95% CI 2-sided [1.59 to 3.40]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0312, Regression, Logistic; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.04 to 2.39]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.40 to 3.19]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.48 to 4.01]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 5]; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 2.39, 95% CI 2-sided [1.45 to 3.94]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0436, Regression, Logistic; Odds Ratio (OR) = 2.10, 95% CI 2-sided [1.02 to 4.32]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority; p = 0.1348, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.84 to 3.69]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.58 to 3.36]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 9]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.46 to 3.09]
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.62 to 3.57]
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 11]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.74 to 3.82]
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.47 to 3.70]
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.45, 95% CI 2-sided [1.55 to 3.89]
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0310, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.07 to 3.82]
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 15]; Test type: Superiority; p = 0.0088, Regression, Logistic; Odds Ratio (OR) = 2.31, 95% CI 2-sided [1.24 to 4.34]
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0360, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.03 to 2.16]
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 17]; Test type: Superiority; p = 0.0039, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.19 to 2.51]
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.43 to 3.13]
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority; p = 0.0040, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.20 to 2.62]
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0175, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.10 to 2.74]
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 21]; Test type: Superiority; p = 0.0065, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.19 to 2.94]
Statistical Analysis 23: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0796, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.94 to 3.23]
Statistical Analysis 24: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 23]; Test type: Superiority; p = 0.0718, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.95 to 3.27]
Statistical Analysis 25: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.36 to 2.96]
Statistical Analysis 26: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.78 to 3.93]
Statistical Analysis 27: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.11, 95% CI 2-sided [1.44 to 3.09]
Statistical Analysis 28: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 27]; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.42 to 3.04]
Statistical Analysis 29: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.41 to 3.23]
Statistical Analysis 30: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 29]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.29, 95% CI 2-sided [1.52 to 3.46]
Statistical Analysis 31: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0113, Regression, Logistic; Odds Ratio (OR) = 2.09, 95% CI 2-sided [1.18 to 3.68]
Statistical Analysis 32: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 31]; Test type: Superiority; p = 0.0064, Regression, Logistic; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.25 to 3.85]
Statistical Analysis 33: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16 >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0200, Regression, Logistic; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.07 to 2.31]
Statistical Analysis 34: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 33]; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.43 to 3.14]
Statistical Analysis 35: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16 >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.34 to 2.87]
Statistical Analysis 36: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0141, Regression, Logistic; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.11 to 2.56]
Statistical Analysis 37: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 36]; Test type: Superiority; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.26 to 2.87]
Statistical Analysis 38: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.2286, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.80 to 2.50]
Statistical Analysis 39: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 13, analysis 38]; Test type: Superiority; p = 0.1808, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.84 to 2.57]
Statistical Analysis 40: Comparison: Placebo vs Tanezumab 2.5/5 mg; Week 16, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.57 to 3.36]

14. Secondary Outcome: Percentage of Participants With Cumulative Percent Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 16
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. Physical function: participant's ability to move around and perform usual activities of daily living. WOMAC physical function subscale: 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint (knee or hip) during past 48 hours, calculated as mean of the scores from 17 individual questions scored on a NRS of 0 (minimum difficulty) to 10 (extreme difficulty),higher scores indicate extreme difficulty/worse physical function. Percentage of participants with cumulative reduction (as percent) (greater than 0 %; >= 10 %, 20 %, 30 %, 40 %, 50 %, 60 %, 70 %, 80 % and 90%; = 100 %) in WOMAC physical function subscale from Baseline to Week 16 were reported. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
percentage of participants
  >=0% | 83.6 | 89.2 | 90.6
  >=10% | 75.4 | 81.0 | 83.3
  >=20% | 63.4 | 72.7 | 76.8
  >=30% | 54.3 | 65.8 | 71.7
  >=40% | 44.8 | 60.2 | 65.7
  >=50% | 36.6 | 54.1 | 57.1
  >=60% | 28.9 | 45.0 | 47.6
  >=70% | 22.8 | 34.2 | 36.1
  >=80% | 15.5 | 24.7 | 26.2
  >=90% | 10.3 | 14.3 | 14.6
  =100% | 2.2 | 6.5 | 7.3

15. Secondary Outcome: Percentage of Participants Achieving Improvement of >=2 Points in Patient's Global Assessment (PGA) of Osteoarthritis
Description: PGA of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, where, 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worse condition. Percentage of participants with improvement of at least 2 points from Baseline in PGA of osteoarthritis were reported. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
percentage of participants
  Week 2 | 19.8 | 25.1 | 22.3
  Week 4 | 20.7 | 27.7 | 27.5
  Week 8 | 24.6 | 26.8 | 27.9
  Week 12 | 26.7 | 34.2 | 39.1
  Week 16 | 22.8 | 30.3 | 31.3
  Week 24: number analyzed (Participants) | 185 | 200 | 202
  Week 24 | 21.1 | 21.0 | 25.7
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline PGA of osteoarthritis, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.1463, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.88 to 2.34]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.9644, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.60 to 1.62]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline PGA of osteoarthritis, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0422, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.02 to 2.59]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 15, analysis 3]; Test type: Superiority; p = 0.1995, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.85 to 2.16]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline PGA of osteoarthritis, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.4878, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.75 to 1.84]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority; p = 0.7856, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.68 to 1.67]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline PGA of osteoarthritis, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0476, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.00 to 2.39]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 15, analysis 7]; Test type: Superiority; p = 0.0124, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.12 to 2.63]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline PGA of osteoarthritis, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0307, Regression, Logistic; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.05 to 2.62]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority; p = 0.0846, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.95 to 2.35]

16. Secondary Outcome: Change From Baseline for Average Pain Score in the Index Joint at Weeks 1, 2, 3, 4, 6, 8, 10, 12 and 16
Description: Participants assessed their average pain in the index hip/knee in the past 24 hours using a scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicated higher pain. Data represents averages of the values reported during the 4-week interval up to and including the given week. Change from baseline was calculated using the difference between each post-baseline weekly mean and the baseline mean score.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 10, 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Change at Week 1 | -1.27 (0.15) | -1.60 (0.15) | -1.65 (0.15)
  Change at Week 2 | -1.68 (0.19) | -2.32 (0.19) | -2.23 (0.19)
  Change at Week 3 | -1.95 (0.20) | -2.61 (0.20) | -2.71 (0.20)
  Change at Week 4 | -1.88 (0.20) | -2.79 (0.20) | -2.82 (0.20)
  Change at Week 6 | -2.17 (0.21) | -2.89 (0.21) | -2.85 (0.21)
  Change at Week 8 | -2.29 (0.21) | -2.73 (0.21) | -2.70 (0.20)
  Change at Week 10 | -2.51 (0.21) | -3.19 (0.21) | -3.19 (0.21)
  Change at Week 12 | -2.58 (0.21) | -3.30 (0.21) | -3.33 (0.21)
  Change at Week 16 | -2.30 (0.22) | -2.98 (0.23) | -3.12 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 1: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0319, ANCOVA; Least Square Mean Difference = -0.33, 95% CI 2-sided [-0.63 to -0.03], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; Week 1:Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0139, ANCOVA; Least Square Mean Difference = -0.38, 95% CI 2-sided [-0.68 to -0.08], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0011, ANCOVA; Least Square Mean Difference = -0.64, 95% CI 2-sided [-1.03 to -0.25], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 16, analysis 3]; Test type: Superiority; p = 0.0053, ANCOVA; Least Square Mean Difference = -0.55, 95% CI 2-sided [-0.93 to -0.16], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 3: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0014, ANCOVA; Least Square Mean Difference = -0.67, 95% CI 2-sided [-1.08 to -0.26], Standard Error of Mean 0.21
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 16, analysis 5]; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean Difference = -0.77, 95% CI 2-sided [-1.17 to -0.36], Standard Error of Mean 0.21
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.91, 95% CI 2-sided [-1.33 to -0.49], Standard Error of Mean 0.22
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.94, 95% CI 2-sided [-1.36 to -0.52], Standard Error of Mean 0.21
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 6: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0015, ANCOVA; Least Square Mean Difference = -0.72, 95% CI 2-sided [-1.16 to -0.28], Standard Error of Mean 0.23
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 16, analysis 9]; Test type: Superiority; p = 0.0023, ANCOVA; Least Square Mean Difference = -0.68, 95% CI 2-sided [-1.12 to -0.24], Standard Error of Mean 0.22
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0512, ANCOVA; Least Square Mean Difference = -0.44, 95% CI 2-sided [-0.89 to 0.00], Standard Error of Mean 0.23
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 16, analysis 11]; Test type: Superiority; p = 0.0693, ANCOVA; Least Square Mean Difference = -0.41, 95% CI 2-sided [-0.85 to 0.03], Standard Error of Mean 0.22
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Week 10: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0043, ANCOVA; Least Square Mean Difference = -0.68, 95% CI 2-sided [-1.14 to -0.21], Standard Error of Mean 0.24
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority; p = 0.0041, ANCOVA; Least Square Mean Difference = -0.67, 95% CI 2-sided [-1.13 to -0.21], Standard Error of Mean 0.23
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0024, ANCOVA; Least Square Mean Difference = -0.73, 95% CI 2-sided [-1.19 to -0.26], Standard Error of Mean 0.24
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 16, analysis 15]; Test type: Superiority; p = 0.0015, ANCOVA; Least Square Mean Difference = -0.75, 95% CI 2-sided [-1.22 to -0.29], Standard Error of Mean 0.24
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline diary average pain as covariate, and study site as a random effect; Test type: Superiority; p = 0.0063, ANCOVA; Least Square Mean Difference = -0.67, 95% CI 2-sided [-1.16 to -0.19], Standard Error of Mean 0.25
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 16, analysis 17]; Test type: Superiority; p = 0.0008, ANCOVA; Least Square Mean Difference = -0.82, 95% CI 2-sided [-1.30 to -0.34], Standard Error of Mean 0.24

17. Secondary Outcome: Change From Baseline for Average Pain Score in the Index Joint at Weeks 20 and 24
Description: Participants assessed their average pain in the index hip/knee in the past 24 hours using a scale ranging from 0 (no pain) to 10 (worst possible pain) weekly beginning at Week 16. Higher scores indicated higher pain. Data represents averages of the values reported during the 4-week interval up to and including the given week. Change from baseline was calculated using the difference between each post-baseline weekly mean and the baseline mean score.
Time Frame: Baseline, Weeks 20 and 24
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either Tanezumab or placebo). Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline: number analyzed (Participants) | 228 | 228 | 231
  Baseline | 7.27 (1.33) | 6.89 (1.63) | 7.13 (1.48)
  Change at Week 20: number analyzed (Participants) | 203 | 209 | 212
  Change at Week 20 | -2.58 (2.34) | -2.76 (2.39) | -3.26 (2.65)
  Change at Week 24: number analyzed (Participants) | 186 | 200 | 197
  Change at Week 24 | -2.63 (2.32) | -2.14 (2.37) | -2.70 (2.69)

18. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Weeks 2, 4, 8, 12 and 16
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. Stiffness was defined as a sensation of decreased ease of movement in the index joint (knee or hip).The WOMAC stiffness subscale was a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in the index joint (knee or hip) during the past 48 hours. It was calculated as mean of the scores from 2 individual questions scored on NRS of 0 (no stiffness) to 10 (extreme stiffness), where higher scores indicated higher stiffness.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Change at Week 2 | -1.85 (0.22) | -2.90 (0.22) | -2.90 (0.21)
  Change at Week 4 | -2.04 (0.22) | -3.28 (0.22) | -3.27 (0.22)
  Change at Week 8 | -2.34 (0.22) | -3.13 (0.22) | -3.08 (0.22)
  Change at Week 12 | -2.55 (0.23) | -3.59 (0.23) | -3.75 (0.23)
  Change at Week 16 | -2.38 (0.23) | -3.22 (0.23) | -3.37 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.04, 95% CI 2-sided [-1.47 to -0.61], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; Least Mean Square Difference = -1.05, 95% CI 2-sided [-1.47 to -0.62], Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.24, 95% CI 2-sided [-1.67 to -0.81], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 18, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.23, 95% CI 2-sided [-1.66 to -0.80], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0007, ANCOVA; Least Square Mean Difference = -0.79, 95% CI 2-sided [-1.25 to -0.33], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 18, analysis 5]; Test type: Superiority; p = 0.0013, ANCOVA; Least Square Mean Difference = -0.74, 95% CI 2-sided [-1.20 to -0.29], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.03, 95% CI 2-sided [-1.51 to -0.55], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 18, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.20, 95% CI 2-sided [-1.67 to -0.73], Standard Error of Mean 0.24
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0007, ANCOVA; Least Square Mean Difference = -0.84, 95% CI 2-sided [-1.32 to -0.35], Standard Error of Mean 0.25
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 18, analysis 9]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.00, 95% CI 2-sided [-1.48 to -0.51], Standard Error of Mean 0.25

19. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Week 24
Description: as for outcome 18
Time Frame: Baseline, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline | 7.49 (1.38) | 7.27 (1.40) | 7.58 (1.40)
  Change at Week 24: number analyzed (Participants) | 185 | 200 | 202
  Change at Week 24 | -2.77 (2.66) | -2.74 (2.70) | -2.86 (2.60)

20. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 2, 4, 8, 12 and 16
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [extreme pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [extreme difficulty], higher score = worse physical function) and WOMAC stiffness subscale assess the amount of stiffness experienced (score: 0 [no stiffness] to 10 [extreme stiffness], higher score = higher stiffness). WOMAC average score was the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 to 10, where higher scores indicated worse response.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Change at Week 2 | -2.07 (0.21) | -2.88 (0.20) | -2.95 (0.20)
  Change at Week 4 | -2.24 (0.21) | -3.28 (0.21) | -3.31 (0.21)
  Change at Week 8 | -2.49 (0.21) | -3.17 (0.21) | -3.08 (0.21)
  Change at Week 12 | -2.70 (0.22) | -3.59 (0.22) | -3.74 (0.22)
  Change at Week 16 | -2.53 (0.22) | -3.22 (0.22) | -3.39 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.82, 95% CI 2-sided [-1.22 to -0.41], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.88, 95% CI 2-sided [-1.29 to -0.48], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.05, 95% CI 2-sided [-1.46 to -0.63], Standard Error of Mean 0.21
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 20, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.07, 95% CI 2-sided [-1.49 to -0.66], Standard Error of Mean 0.21
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0024, ANCOVA; Least Square Mean Difference = -0.68, 95% CI 2-sided [-1.12 to -0.24], Standard Error of Mean 0.22
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 20, analysis 5]; Test type: Superiority; p = 0.0078, ANCOVA; Least Square Mean Difference = -0.59, 95% CI 2-sided [-1.03 to -0.16], Standard Error of Mean 0.22
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean Difference = -0.89, 95% CI 2-sided [-1.35 to -0.43], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 20, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.04, 95% CI 2-sided [-1.50 to -0.57], Standard Error of Mean 0.24
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0034, ANCOVA; Least Square Mean Difference = -0.70, 95% CI 2-sided [-1.16 to -0.23], Standard Error of Mean 0.24
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 20, analysis 9]; Test type: Superiority; p = 0.0003, ANCOVA; Least Square Mean Difference = -0.87, 95% CI 2-sided [-1.33 to -0.40], Standard Error of Mean 0.24

21. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 24
Description: as for outcome 20
Time Frame: Baseline, Week 24
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either Tanezumab or placebo).Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline | 7.39 (1.11) | 7.18 (1.11) | 7.44 (1.17)
  Change at Week 24: number analyzed (Participants) | 185 | 200 | 202
  Change at Week 24 | -2.96 (2.37) | -2.80 (2.48) | -2.94 (2.41)

22. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item (Pain When Walking on a Flat Surface) at Weeks 2, 4, 8, 12 and 16
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis in index joint (knee or hip). Participants answered a question: "How much pain have you had when walking on a flat surface?". Participants responded about the amount of pain they experienced when walking on a flat surface by using a NRS of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Change at Week 2 | -2.09 (0.21) | -2.75 (0.21) | -2.76 (0.21)
  Change at Week 4 | -2.31 (0.21) | -3.16 (0.21) | -3.22 (0.21)
  Change at Week 8 | -2.55 (0.21) | -3.19 (0.21) | -2.89 (0.21)
  Change at Week 12 | -2.77 (0.23) | -3.53 (0.23) | -3.60 (0.23)
  Change at Week 16 | -2.57 (0.23) | -3.17 (0.23) | -3.24 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects,baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0026, ANCOVA; Least Square Mean Difference = -0.66, 95% CI 2-sided [-1.10 to -0.23], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.0023, ANCOVA; Least Mean Square Difference = -0.67, 95% CI 2-sided [-1.10 to -0.24], Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects,baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean Difference = -0.85, 95% CI 2-sided [-1.29 to -0.40], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 22, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.91, 95% CI 2-sided [-1.35 to -0.47], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects,baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0066, ANCOVA; Least Square Mean Difference = -0.64, 95% CI 2-sided [-1.11 to -0.18], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 22, analysis 5]; Test type: Superiority; p = 0.1506, ANCOVA; Least Square Mean Difference = -0.34, 95% CI 2-sided [-0.79 to 0.12], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects,baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0021, ANCOVA; Least Square Mean Difference = -0.76, 95% CI 2-sided [-1.25 to -0.28], Standard Error of Mean 0.25
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p = 0.0008, ANCOVA; Least Square Mean Difference = -0.83, 95% CI 2-sided [-1.32 to -0.35], Standard Error of Mean 0.25
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects,baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0167, ANCOVA; Least Square Mean Difference = -0.60, 95% CI 2-sided [-1.09 to -0.11], Standard Error of Mean 0.25
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 22, analysis 9]; Test type: Superiority; p = 0.0073, ANCOVA; Least Square Mean Difference = -0.68, 95% CI 2-sided [-1.17 to -0.18], Standard Error of Mean 0.25

23. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item (Pain When Walking on a Flat Surface) at Week 24
Description: as for outcome 22
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline | 7.22 (1.39) | 7.03 (1.40) | 7.24 (1.42)
  Change at Week 24: number analyzed (Participants) | 185 | 200 | 202
  Change at Week 24 | -2.93 (2.71) | -2.64 (2.69) | -2.74 (2.72)

24. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale (Pain When Going up or Down Stairs) at Weeks 2, 4, 8, 12 and 16
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis in index joint (knee or hip). Participants answered a question: "How much pain have you had when going up or down the stairs?" Participants responded about the amount of pain they experienced when going up or down stairs by using a NRS of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Change at Week 2 | -2.24 (0.22) | -2.88 (0.22) | -3.10 (0.22)
  Change at Week 4 | -2.53 (0.23) | -3.50 (0.23) | -3.63 (0.22)
  Change at Week 8 | -2.77 (0.22) | -3.40 (0.22) | -3.21 (0.22)
  Change at Week 12 | -2.97 (0.24) | -3.82 (0.24) | -3.94 (0.23)
  Change at Week 16 | -2.70 (0.24) | -3.40 (0.24) | -3.59 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0058, ANCOVA; Least Square Mean Difference = -0.64, 95% CI 2-sided [-1.09 to -0.18], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean Difference = -0.86, 95% CI 2-sided [-1.31 to -0.41], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.98, 95% CI 2-sided [-1.44 to -0.51], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 24, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.10, 95% CI 2-sided [-1.56 to -0.64], Standard Error of Mean 0.23
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0091, ANCOVA; Least Square Mean Difference = -0.63, 95% CI 2-sided [-1.11 to -0.16], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 24, analysis 5]; Test type: Superiority; p = 0.0668, ANCOVA; Least Square Mean Difference = -0.44, 95% CI 2-sided [-0.92 to 0.03], Standard Error of Mean 0.24
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0011, ANCOVA; Least Square Mean Difference = -0.85, 95% CI 2-sided [-1.36 to -0.34], Standard Error of Mean 0.26
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 24, analysis 7]; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean Difference = -0.97, 95% CI 2-sided [-1.48 to -0.46], Standard Error of Mean 0.26
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0059, ANCOVA; Least Square Mean Difference = -0.70, 95% CI 2-sided [-1.20 to -0.20], Standard Error of Mean 0.25
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 24, analysis 9]; Test type: Superiority; p = 0.0005, ANCOVA; Least Square Mean Difference = -0.89, 95% CI 2-sided [-1.39 to -0.39], Standard Error of Mean 0.25

25. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale (Pain When Going up or Down Stairs) at Week 24
Description: as for outcome 24
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline | 8.09 (1.23) | 7.91 (1.22) | 8.13 (1.24)
  Change at Week 24: number analyzed (Participants) | 185 | 200 | 202
  Change at Week 24 | -3.12 (2.62) | -2.76 (2.52) | -2.86 (2.65)

26. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire for Osteoarthritis (WPAI:OA) Scores at Baseline
Description: WPAI is 6-question participant rated questionnaire to determine the impact of osteoarthritis on absenteeism, presenteeism, work productivity, and daily activity impairment for a period of 7 days prior to a visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism), overall work impairment (work productivity) and activity impairment (daily activity impairment). These sub-scores are expressed as an impairment percentage (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either Tanezumab or placebo). Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Percent Work Time Missed: number analyzed (Participants) | 88 | 100 | 94
  Percent Work Time Missed | 4.6 (12.96) | 7.4 (17.42) | 8.4 (18.15)
  Percent Impairment While Working: number analyzed (Participants) | 88 | 100 | 93
  Percent Impairment While Working | 60.9 (19.51) | 59.5 (21.57) | 60.1 (21.39)
  Percent Overall Work Impairment: number analyzed (Participants) | 88 | 100 | 93
  Percent Overall Work Impairment | 62.3 (20.42) | 61.8 (22.28) | 62.0 (21.61)
  Percent Activity Impairment | 69.4 (14.62) | 68.3 (15.56) | 69.8 (16.00)

27. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire for Osteoarthritis (WPAI:OA) Scores at Week 16
Description: as for outcome 26
Time Frame: Baseline and Week 16
Population: as for outcome 26
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Change at Week 16: Percent Work Time Missed: number analyzed (Participants) | 63 | 83 | 75
  Change at Week 16: Percent Work Time Missed | -3.58 (1.27) | -2.97 (1.17) | -5.26 (1.23)
  Change at Week 16:Percent Impairment While Working: number analyzed (Participants) | 63 | 82 | 75
  Change at Week 16:Percent Impairment While Working | -21.89 (3.46) | -27.32 (3.24) | -27.48 (3.39)
  Change at Week 16: Percent Overall Work Impairment: number analyzed (Participants) | 63 | 82 | 75
  Change at Week 16: Percent Overall Work Impairment | -22.48 (3.52) | -28.28 (3.29) | -28.87 (3.44)
  Change at Week 16: Percent Activity Impairment: number analyzed (Participants) | 194 | 215 | 212
  Change at Week 16: Percent Activity Impairment | -26.72 (2.18) | -30.55 (2.16) | -30.49 (2.14)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Percent Work Time Missed: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.6984, ANCOVA; Least Square Mean Difference = 0.61, 95% CI 2-sided [-2.48 to 3.70], Standard Error of Mean 1.56
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority; p = 0.2953, ANCOVA; Least Square Mean Difference = -1.68, 95% CI 2-sided [-4.84 to 1.48], Standard Error of Mean 1.60
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Percent Impairment While Working: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.1911, ANCOVA; Least Square Mean Difference = -5.43, 95% CI 2-sided [-13.59 to 2.74], Standard Error of Mean 4.14
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 27, analysis 3]; Test type: Superiority; p = 0.1857, ANCOVA; Least Square Mean Difference = -5.59, 95% CI 2-sided [-13.89 to 2.71], Standard Error of Mean 4.20
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Percent Overall Work Impairment: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.1707, ANCOVA; Least Square Mean Difference = -5.80, 95% CI 2-sided [-14.12 to 2.52], Standard Error of Mean 4.21
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 27, analysis 5]; Test type: Superiority; p = 0.1380, ANCOVA; Least Square Mean Difference = -6.39, 95% CI 2-sided [-14.85 to 2.07], Standard Error of Mean 4.29
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Percent Activity Impairment: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.1151, ANCOVA; Least Square Mean Difference = -3.82, 95% CI 2-sided [-8.58 to 0.94], Standard Error of Mean 2.42
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 27, analysis 7]; Test type: Superiority; p = 0.1195, ANCOVA; Least Square Mean Difference = -3.77, 95% CI 2-sided [-8.51 to 0.98], Standard Error of Mean 2.41

28. Secondary Outcome: European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Dimensions Score
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The health utility score for a patient with no problems in all 5 items is 1 for all countries (except for Zimbabwe where it is 0.9), and is reduced where a patient reports greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8 and 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline: Mobility | 3.0 (0.71) | 3.0 (0.68) | 3.0 (0.63)
  Baseline: Self-care | 2.2 (0.90) | 2.3 (0.90) | 2.3 (0.88)
  Baseline: Usual activities | 2.9 (0.74) | 3.0 (0.72) | 3.0 (0.73)
  Baseline: Pain/Discomfort | 3.3 (0.73) | 3.4 (0.68) | 3.4 (0.73)
  Baseline: Anxiety/Depression | 1.5 (0.77) | 1.5 (0.77) | 1.6 (0.87)
  Week 8: Mobility: number analyzed (Participants) | 222 | 228 | 224
  Week 8: Mobility | 2.3 (0.84) | 2.1 (0.86) | 2.2 (0.84)
  Week 8: Self-care: number analyzed (Participants) | 222 | 228 | 224
  Week 8: Self-care | 1.6 (0.78) | 1.5 (0.76) | 1.6 (0.79)
  Week 8: Usual activities: number analyzed (Participants) | 222 | 228 | 224
  Week 8: Usual activities | 2.2 (0.85) | 2.1 (0.84) | 2.1 (0.83)
  Week 8: Pain/Discomfort: number analyzed (Participants) | 222 | 228 | 224
  Week 8: Pain/Discomfort | 2.6 (0.78) | 2.4 (0.80) | 2.4 (0.85)
  Week 8: Anxiety/Depression: number analyzed (Participants) | 222 | 228 | 224
  Week 8: Anxiety/Depression | 1.4 (0.67) | 1.3 (0.56) | 1.4 (0.65)
  Week 16: Mobility: number analyzed (Participants) | 194 | 215 | 211
  Week 16: Mobility | 2.2 (0.89) | 2.1 (0.85) | 2.0 (0.89)
  Week 16: Self-care: number analyzed (Participants) | 194 | 215 | 211
  Week 16: Self-care | 1.6 (0.77) | 1.6 (0.78) | 1.5 (0.70)
  Week 16: Usual activities: number analyzed (Participants) | 194 | 215 | 211
  Week 16: Usual activities | 2.1 (0.91) | 2.0 (0.86) | 2.0 (0.88)
  Week 16: Pain/Discomfort: number analyzed (Participants) | 194 | 215 | 211
  Week 16: Pain/Discomfort | 2.4 (0.87) | 2.3 (0.81) | 2.3 (0.92)
  Week 16: Anxiety/Depression: number analyzed (Participants) | 194 | 215 | 211
  Week 16: Anxiety/Depression | 1.4 (0.66) | 1.3 (0.62) | 1.3 (0.64)

29. Secondary Outcome: European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Overall Health Utility Score/Index Value
Description: EQ-5D-5L: standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional VAS. EQ-5D health state profile comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Responses from the five domains were used to calculate a single utility index (the Overall health utility score) where values are <=1. The Overall health utility score for a patient with no problems in all 5 items is 1 for all countries (except for Zimbabwe where it is 0.9), and is reduced where a patient reports greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8 and 16
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline | 0.63 (0.14) | 0.63 (0.13) | 0.61 (0.14)
  Week 8: number analyzed (Participants) | 222 | 228 | 224
  Week 8 | 0.75 (0.12) | 0.77 (0.12) | 0.76 (0.13)
  Week 16: number analyzed (Participants) | 194 | 215 | 211
  Week 16 | 0.76 (0.13) | 0.77 (0.13) | 0.78 (0.14)

30. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits of Services Directly Related to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 40) and past 8 weeks (for Week 24). Visits of services directly related to osteoarthritis evaluated were: visits to primary care physician, neurologist, rheumatologist, physician assistant or nurse practitioner, pain specialist, orthopedist, physical therapist, chiropractor, alternative medicine or therapy, podiatrist, nutritionist/dietitian, radiologist, home healthcare services and other practitioner.
Time Frame: Baseline, Weeks 24 and 40
Population: as for outcome 26
Measure: Median (Full Range); unit: visits
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
visits
  Baseline:Primary Care Physician: number analyzed (Participants) | 117 | 106 | 111
  Baseline:Primary Care Physician | 1.0 [1.0 to 190.0] | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 101.0]
  Baseline: Neurologist: number analyzed (Participants) | 1 | 3 | 1
  Baseline: Neurologist | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]
  Baseline: Rheumatologist: number analyzed (Participants) | 6 | 3 | 10
  Baseline: Rheumatologist | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 4.0]
  Baseline:Physician assistant or nurse practitioner: number analyzed (Participants) | 8 | 11 | 9
  Baseline:Physician assistant or nurse practitioner | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 2.0]
  Baseline:Pain specialist: number analyzed (Participants) | 9 | 7 | 11
  Baseline:Pain specialist | 2.0 [1.0 to 10.0] | 3.0 [1.0 to 190.0] | 1.0 [1.0 to 21.0]
  Baseline: Orthopedist: number analyzed (Participants) | 19 | 28 | 27
  Baseline: Orthopedist | 1.0 [1.0 to 90.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 3.0]
  Baseline: Physical therapist: number analyzed (Participants) | 16 | 14 | 17
  Baseline: Physical therapist | 3.0 [1.0 to 24.0] | 2.0 [1.0 to 14.0] | 3.0 [1.0 to 60.0]
  Baseline:Chiropractor: number analyzed (Participants) | 10 | 12 | 13
  Baseline:Chiropractor | 2.0 [1.0 to 6.0] | 3.0 [1.0 to 10.0] | 4.0 [1.0 to 120.0]
  Baseline:Alternative medicine or therapy: number analyzed (Participants) | 11 | 15 | 17
  Baseline:Alternative medicine or therapy | 2.0 [1.0 to 90.0] | 2.0 [1.0 to 10.0] | 2.0 [1.0 to 8.0]
  Baseline:Podiatrist: number analyzed (Participants) | 1 | 4 | 4
  Baseline:Podiatrist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Baseline:Nutritionist/Dietitian: number analyzed (Participants) | 5 | 5 | 3
  Baseline:Nutritionist/Dietitian | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0]
  Baseline:Radiologist: number analyzed (Participants) | 26 | 22 | 17
  Baseline:Radiologist | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 4.0]
  Baseline:Home healthcare services: number analyzed (Participants) | 1 | 1 | 3
  Baseline:Home healthcare services | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0] | 2.0 [1.0 to 7.0]
  Baseline: Other Practitioner: number analyzed (Participants) | 19 | 17 | 18
  Baseline: Other Practitioner | 1.0 [1.0 to 90.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 120.0]
  Week 24:Primary Care Physician: number analyzed (Participants) | 42 | 48 | 53
  Week 24:Primary Care Physician | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 3.0]
  Week 24: Neurologist: number analyzed (Participants) | 0 | 2 | 0
  Week 24: Neurologist |  | 1.0 [1.0 to 1.0] |
  Week 24: Rheumatologist: number analyzed (Participants) | 6 | 4 | 3
  Week 24: Rheumatologist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Week 24: Physician Assistant Or Nurse Practitioner: number analyzed (Participants) | 3 | 0 | 1
  Week 24: Physician Assistant Or Nurse Practitioner | 1.0 [1.0 to 1.0] |  | 2.0 [2.0 to 2.0]
  Week 24: Pain Specialist: number analyzed (Participants) | 5 | 4 | 2
  Week 24: Pain Specialist | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Week 24: Orthopedist: number analyzed (Participants) | 11 | 13 | 11
  Week 24: Orthopedist | 1.0 [1.0 to 101.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0]
  Week 24: Physical Therapist: number analyzed (Participants) | 8 | 7 | 7
  Week 24: Physical Therapist | 2.5 [1.0 to 5.0] | 2.0 [1.0 to 11.0] | 8.0 [1.0 to 20.0]
  Week 24: Chiropractor: number analyzed (Participants) | 6 | 3 | 6
  Week 24: Chiropractor | 2.0 [1.0 to 16.0] | 1.0 [1.0 to 2.0] | 2.5 [2.0 to 4.0]
  Week 24: Alternative Medicine Or Therapy: number analyzed (Participants) | 4 | 4 | 4
  Week 24: Alternative Medicine Or Therapy | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 8.0]
  Week 24: Podiatrist: number analyzed (Participants) | 2 | 2 | 1
  Week 24: Podiatrist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Week 24: Nutritionist/Dietitian: number analyzed (Participants) | 2 | 4 | 1
  Week 24: Nutritionist/Dietitian | 2.5 [2.0 to 3.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Week 24: Radiologist: number analyzed (Participants) | 4 | 5 | 3
  Week 24: Radiologist | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Week 24: Other Practitioner: number analyzed (Participants) | 10 | 7 | 13
  Week 24: Other Practitioner | 1.0 [1.0 to 110.0] | 2.0 [1.0 to 190.0] | 1.0 [1.0 to 6.0]
  Week 40: Primary Care Physician: number analyzed (Participants) | 49 | 54 | 58
  Week 40: Primary Care Physician | 1.0 [1.0 to 11.0] | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 101.0]
  Week 40: Neurologist: number analyzed (Participants) | 1 | 1 | 1
  Week 40: Neurologist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Week 40: Rheumatologist: number analyzed (Participants) | 2 | 5 | 2
  Week 40: Rheumatologist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Week 40: Physician Assistant Or Nurse Practitioner: number analyzed (Participants) | 3 | 6 | 5
  Week 40: Physician Assistant Or Nurse Practitioner | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 111.0]
  Week 40: Pain Specialist: number analyzed (Participants) | 4 | 10 | 5
  Week 40: Pain Specialist | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 111.0] | 2.0 [1.0 to 5.0]
  Week 40: Orthopedist: number analyzed (Participants) | 12 | 14 | 19
  Week 40: Orthopedist | 1.5 [1.0 to 190.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 101.0]
  Week 40: Physical Therapist: number analyzed (Participants) | 9 | 9 | 1
  Week 40: Physical Therapist | 8.0 [1.0 to 12.0] | 6.0 [1.0 to 10.0] | 4.0 [4.0 to 4.0]
  Week 40: Chiropractor: number analyzed (Participants) | 6 | 6 | 5
  Week 40: Chiropractor | 1.0 [1.0 to 4.0] | 3.0 [1.0 to 4.0] | 5.0 [1.0 to 16.0]
  Week 40: Alternative Medicine Or Therapy: number analyzed (Participants) | 6 | 6 | 4
  Week 40: Alternative Medicine Or Therapy | 3.0 [1.0 to 6.0] | 1.5 [1.0 to 9.0] | 2.5 [1.0 to 111.0]
  Week 40: Podiatrist: number analyzed (Participants) | 1 | 2 | 2
  Week 40: Podiatrist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Week 40: Nutritionist/Dietitian: number analyzed (Participants) | 0 | 2 | 2
  Week 40: Nutritionist/Dietitian |  | 3.5 [1.0 to 6.0] | 1.5 [1.0 to 2.0]
  Week 40: Radiologist: number analyzed (Participants) | 5 | 6 | 10
  Week 40: Radiologist | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Week 40: Home Healthcare Services: number analyzed (Participants) | 1 | 1 | 4
  Week 40: Home Healthcare Services | 1.0 [1.0 to 1.0] | 30.0 [30.0 to 30.0] | 7.5 [3.0 to 11.0]
  Week 40: Other Practitioner: number analyzed (Participants) | 6 | 8 | 9
  Week 40: Other Practitioner | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 111.0]

31. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Visited the Emergency Room Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 40) and past 8 weeks (for Week 24). Domain evaluated was number of participants who visited the emergency room due to osteoarthritis (OA).
Time Frame: Baseline, Weeks 24 and 40
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
Participants
  Baseline | 1 | 2 | 4
  Week 24: number analyzed (Participants) | 196 | 202 | 206
  Week 24 | 0 | 0 | 2
  Week 40: number analyzed (Participants) | 184 | 194 | 192
  Week 40 | 2 | 1 | 1

32. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits to the Emergency Room Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 40) and past 8 weeks (for Week 24). Domain evaluated was number of visits to the emergency room due to OA.
Time Frame: Baseline, Weeks 24 and 40
Population: as for outcome 17
Measure: Median (Full Range); unit: visits
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
visits
  Baseline: number analyzed (Participants) | 1 | 2 | 4
  Baseline | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]
  Week 24: number analyzed (Participants) | 0 | 0 | 2
  Week 24 |  |  | 2.5 [1.0 to 4.0]
  Week 40: number analyzed (Participants) | 2 | 1 | 1
  Week 40 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

33. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Hospitalized Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 40) and past 8 weeks (for Week 24). Domain evaluated was number of participants who were hospitalized due to OA.
Time Frame: Baseline, Weeks 24 and 40
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
Participants
  Baseline | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 196 | 202 | 206
  Week 24 | 2 | 0 | 2
  Week 40: number analyzed (Participants) | 184 | 194 | 192
  Week 40 | 2 | 0 | 2

34. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Nights Stayed in the Hospital Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 40) and past 8 weeks (for Week 24). Domain evaluated was number of nights stayed in the hospital due to OA.
Time Frame: Baseline, Weeks 24 and 40
Population: as for outcome 17
Measure: Median (Full Range); unit: nights
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
nights
  Baseline: number analyzed (Participants) | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 2 | 0 | 2
  Week 24 | 3.0 [2.0 to 4.0] |  | 2.0 [1.0 to 3.0]
  Week 40: number analyzed (Participants) | 2 | 0 | 2
  Week 40 | 3.5 [3.0 to 4.0] |  | 1.5 [1.0 to 2.0]

35. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Used Any Aids/Devices for Doing Things
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 40) and past 8 weeks (for Week 24). Domain evaluated was number of participants who used any aids/devices for doing things. Aids such as walking aid, wheelchair, device or utensil for dress/bathe/eat and any other aids/devices.
Time Frame: Baseline, Weeks 24 and 40
Population: The intent to treat (ITT) population included all randomized participants who received at least one dose of subcutaneous (SC) study medication (either Tanezumab or placebo). Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
Participants
  Baseline:Walking Aid Use: Never | 196 | 187 | 189
  Baseline:Walking Aid Use: Rarely | 2 | 5 | 10
  Baseline:Walking Aid Use: Sometimes | 18 | 23 | 15
  Baseline:Walking Aid Use: Often | 11 | 10 | 13
  Baseline:Walking Aid Use: Always | 5 | 6 | 6
  Baseline:Wheelchair Use: Never | 229 | 230 | 230
  Baseline:Wheelchair Use: Rarely | 2 | 1 | 0
  Baseline:Wheelchair Use: Sometimes | 1 | 0 | 2
  Baseline:Wheelchair Use: Often | 0 | 0 | 1
  Baseline:Wheelchair Use: Always | 0 | 0 | 0
  Baseline:Device/Utensil to Dress Bathe Eat: Never | 228 | 221 | 225
  Baseline:Device/Utensil to Dress Bathe Eat: Rarely | 1 | 1 | 1
  Baseline:Device/Utensil to Dress Bathe Eat: Sometimes | 2 | 2 | 4
  Baseline:Device/Utensil to Dress Bathe Eat: Often | 0 | 7 | 2
  Baseline:Device/Utensil to Dress Bathe Eat: Always | 1 | 0 | 1
  Baseline:Other Aids Or Devices:Never: Never | 217 | 211 | 208
  Baseline:Other Aids Or Devices:Never: Rarely | 1 | 4 | 1
  Baseline:Other Aids Or Devices:Never: Sometimes | 4 | 7 | 14
  Baseline:Other Aids Or Devices:Never: Often | 5 | 5 | 6
  Baseline:Other Aids Or Devices:Never: Always | 5 | 4 | 4
  Week 24 :Walking Aid Use:Never: number analyzed (Participants) | 196 | 202 | 206
  Week 24 :Walking Aid Use:Never: Never | 168 | 185 | 175
  Week 24 :Walking Aid Use:Never: Rarely | 6 | 2 | 9
  Week 24 :Walking Aid Use:Never: Sometimes | 11 | 6 | 10
  Week 24 :Walking Aid Use:Never: Often | 4 | 4 | 5
  Week 24 :Walking Aid Use:Never: Always | 7 | 5 | 7
  Week 24:Wheelchair Use:Never: number analyzed (Participants) | 196 | 202 | 206
  Week 24:Wheelchair Use:Never: Never | 195 | 200 | 204
  Week 24:Wheelchair Use:Never: Rarely | 0 | 1 | 0
  Week 24:Wheelchair Use:Never: Sometimes | 1 | 1 | 2
  Week 24:Wheelchair Use:Never: Often | 0 | 0 | 0
  Week 24:Wheelchair Use:Never: Always | 0 | 0 | 0
  Week 24:Device/Utensil-Dress Bathe Eat: number analyzed (Participants) | 196 | 202 | 206
  Week 24:Device/Utensil-Dress Bathe Eat: Never | 195 | 200 | 203
  Week 24:Device/Utensil-Dress Bathe Eat: Rarely | 0 | 0 | 0
  Week 24:Device/Utensil-Dress Bathe Eat: Sometimes | 1 | 1 | 0
  Week 24:Device/Utensil-Dress Bathe Eat: Often | 0 | 0 | 2
  Week 24:Device/Utensil-Dress Bathe Eat: Always | 0 | 1 | 1
  Week 24:Other Aids Or Devices:Never: number analyzed (Participants) | 196 | 202 | 206
  Week 24:Other Aids Or Devices:Never: Never | 189 | 197 | 199
  Week 24:Other Aids Or Devices:Never: Rarely | 2 | 0 | 2
  Week 24:Other Aids Or Devices:Never: Sometimes | 2 | 3 | 2
  Week 24:Other Aids Or Devices:Never: Often | 2 | 2 | 1
  Week 24:Other Aids Or Devices:Never: Always | 1 | 0 | 2
  Week 40 :Walking Aid Use:Never: number analyzed (Participants) | 184 | 194 | 192
  Week 40 :Walking Aid Use:Never: Never | 164 | 175 | 170
  Week 40 :Walking Aid Use:Never: Rarely | 0 | 5 | 2
  Week 40 :Walking Aid Use:Never: Sometimes | 13 | 5 | 7
  Week 40 :Walking Aid Use:Never: Often | 3 | 2 | 6
  Week 40 :Walking Aid Use:Never: Always | 4 | 7 | 7
  Week 40 :Wheelchair Use:Never: number analyzed (Participants) | 184 | 194 | 192
  Week 40 :Wheelchair Use:Never: Never | 183 | 194 | 189
  Week 40 :Wheelchair Use:Never: Rarely | 0 | 0 | 1
  Week 40 :Wheelchair Use:Never: Sometimes | 0 | 0 | 1
  Week 40 :Wheelchair Use:Never: Often | 1 | 0 | 1
  Week 40 :Wheelchair Use:Never: Always | 0 | 0 | 0
  Week 40:Device/Utensil to Dress Bathe Eat: number analyzed (Participants) | 184 | 194 | 192
  Week 40:Device/Utensil to Dress Bathe Eat: Never | 183 | 191 | 188
  Week 40:Device/Utensil to Dress Bathe Eat: Rarely | 0 | 0 | 1
  Week 40:Device/Utensil to Dress Bathe Eat: Sometimes | 0 | 1 | 1
  Week 40:Device/Utensil to Dress Bathe Eat: Often | 0 | 1 | 1
  Week 40:Device/Utensil to Dress Bathe Eat: Always | 1 | 1 | 1
  Week 40:Other Aids Or Devices:Never: number analyzed (Participants) | 184 | 194 | 192
  Week 40:Other Aids Or Devices:Never: Never | 180 | 187 | 187
  Week 40:Other Aids Or Devices:Never: Rarely | 1 | 0 | 2
  Week 40:Other Aids Or Devices:Never: Sometimes | 1 | 1 | 2
  Week 40:Other Aids Or Devices:Never: Often | 1 | 4 | 1
  Week 40:Other Aids Or Devices:Never: Always | 1 | 2 | 0

36. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Quit Job Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage (during 3 months prior to baseline) at baseline, Week 24 and Week 40. Domain evaluated was number of participants who quit job due to OA.
Time Frame: Baseline, Weeks 24 and 40
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
Participants
  Baseline | 7 | 9 | 11
  Week 24: number analyzed (Participants) | 196 | 202 | 206
  Week 24 | 2 | 1 | 5
  Week 40: number analyzed (Participants) | 184 | 194 | 192
  Week 40 | 4 | 6 | 8

37. Secondary Outcome: Health Care Resource Utilization (HCRU): Duration Since Quitting Job Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage (during 3 months prior to baseline) at baseline, Week 24 and Week 40. Domain evaluated was duration since quitting job due to OA.
Time Frame: Baseline, Weeks 24 and 40
Population: ITT population: all randomized participants who received at least one dose of SC study medication (either Tanezumab or placebo). One additional participant apart from the ones who had responded for quitting job responded to duration since quitting job. 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Median (Full Range); unit: years
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
years
  Baseline: number analyzed (Participants) | 7 | 10 | 11
  Baseline | 4.3 [1.6 to 12.0] | 2.2 [0.1 to 14.0] | 4.3 [0.2 to 18.8]
  Week 24: number analyzed (Participants) | 2 | 1 | 5
  Week 24 | 0.9 [0.6 to 1.3] | 5.0 [5.0 to 5.0] | 1.3 [0.1 to 3.1]
  Week 40: number analyzed (Participants) | 4 | 6 | 8
  Week 40 | 1.1 [0.2 to 4.3] | 3.3 [0.2 to 13.1] | 2.5 [0.1 to 13.8]

38. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy
Description: Number of participants who withdrew from treatment due to lack of efficacy have been reported here.
Time Frame: Baseline up to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
Participants | 13 | 6 | 4
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.1444, Regression, Logistic; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.18 to 1.29]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p = 0.0335, Regression, Logistic; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.09 to 0.91]

39. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Time to discontinuation due to lack of efficacy was defined as the time interval from the date of first study drug administration up to the date of discontinuation of participant from treatment due to lack of efficacy.
Time Frame: Baseline up to Week 16
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either Tanezumab or placebo). Here, 'Overall number of participants analyzed' signifies participants who discontinued from the study due to lack of efficacy.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 13 | 6 | 4
days | NA [6 to NA] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy, median and upper limit could not be calculated. | NA [53 to NA] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy, median and upper limit could not be calculated. | NA [43 to NA] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy, median and upper limit could not be calculated.
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Missing data for the selected percentile(s) was due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy; Test type: Superiority; p = 0.0809, Log Rank — P-value was based on the log-rank test
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 39, analysis 1]; Test type: Superiority; p = 0.0239, Log Rank — P-value was based on the log-rank test

40. Secondary Outcome: Number of Participants Who Took Rescue Medication During Weeks 2, 4, 8, 12 and 16
Description: In case of inadequate pain relief, acetaminophen up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between day 1 and week 16. Number of participants with any use of rescue medication during the particular study week were summarized.
Time Frame: Week 2, 4, 8, 12 and 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
Participants
  Week 2: number analyzed (Participants) | 232 | 230 | 233
  Week 2 | 160 | 137 | 138
  Week 4 | 143 | 119 | 110
  Week 8 | 117 | 110 | 117
  Week 12 | 103 | 93 | 88
  Week 16 | 100 | 101 | 96
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0761, Regression, Logistic; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.48 to 1.04]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 40, analysis 1]; Test type: Superiority; p = 0.0312, Regression, Logistic; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.44 to 0.96]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0262, Regression, Logistic; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.45 to 0.95]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 40, analysis 3]; Test type: Superiority; p = 0.0013, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.37 to 0.79]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.6706, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.64 to 1.33]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 40, analysis 5]; Test type: Superiority; p = 0.9720, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.69 to 1.43]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.5311, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.61 to 1.29]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 40, analysis 7]; Test type: Superiority; p = 0.1712, Regression, Logistic; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.53 to 1.12]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.7475, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.73 to 1.54]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 40, analysis 9]; Test type: Superiority; p = 0.6564, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.63 to 1.33]

41. Secondary Outcome: Number of Participants Who Took Rescue Medication During Week 24
Description: In case of inadequate pain relief, after Week 16, acetaminophen up to 3000 mg per day up to 7 days in a week could be taken as rescue medication and use was reported weekly via diary. Number of participants with any use of rescue medication during the 4 weeks up to the particular study week were summarized.
Time Frame: Week 24
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either Tanezumab or placebo). Here, 'Overall number of participants analyzed' signifies participants who took rescue medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 189 | 202 | 199
Participants | 108 | 125 | 118

42. Secondary Outcome: Number of Days of Rescue Medication Use at Week 2, 4, 8, 12 and 16
Description: In case of inadequate pain relief during the treatment period, acetaminophen up to 3000 mg per day up to 3 days in a week could be taken as rescue medication. Number of days the participants used the rescue medication during the particular study weeks were summarized.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
days
  Week 2 | 2.46 (0.24) | 2.27 (0.22) | 2.02 (0.19)
  Week 4 | 2.20 (0.25) | 1.93 (0.22) | 1.68 (0.19)
  Week 8 | 1.77 (0.21) | 1.68 (0.20) | 1.53 (0.18)
  Week 12 | 1.45 (0.21) | 1.31 (0.18) | 1.12 (0.16)
  Week 16 | 1.48 (0.22) | 1.57 (0.21) | 1.39 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.4833, Negative binomial model; LS Mean Ratio = 0.92, 95% CI 2-sided [0.73 to 1.16], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; Test type: Superiority — Week 2: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; p = 0.0942, Negative binomial model; LS Mean Ratio = 0.82, 95% CI 2-sided [0.65 to 1.03], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.3371, Negative binomial model; LS Mean Ratio = 0.88, 95% CI 2-sided [0.67 to 1.15], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 42, analysis 3]; Test type: Superiority; p = 0.0508, Negative binomial model; LS Mean Ratio = 0.76, 95% CI 2-sided [0.58 to 1.00], Standard Error of Mean 0.11
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.7280, Negative binomial model; LS Mean Ratio = 0.95, 95% CI 2-sided [0.71 to 1.27], Standard Error of Mean 0.14
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 42, analysis 5]; Test type: Superiority; p = 0.3244, Negative binomial model; LS Mean Ratio = 0.87, 95% CI 2-sided [0.65 to 1.15], Standard Error of Mean 0.13
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.5681, Negative binomial model; LS Mean Ratio = 0.91, 95% CI 2-sided [0.65 to 1.27], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 42, analysis 7]; Test type: Superiority; p = 0.1387, Negative binomial model; LS Mean Ratio = 0.77, 95% CI 2-sided [0.55 to 1.09], Standard Error of Mean 0.13
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.7275, Negative binomial model; LS Mean Ratio = 1.06, 95% CI 2-sided [0.76 to 1.48], Standard Error of Mean 0.18
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 42, analysis 9]; Test type: Superiority; p = 0.7090, Negative binomial model; LS Mean Ratio = 0.94, 95% CI 2-sided [0.67 to 1.31], Standard Error of Mean 0.16

43. Secondary Outcome: Number of Days of Rescue Medication Use at Week 24
Description: In case of inadequate pain relief, after Week 16, acetaminophen up to 3000 mg per day up to 7 days in a week could be taken as rescue medication and use was reported weekly via diary. Number of days per week the participants used the rescue medication during the 4 weeks up to the particular study week were summarized.
Time Frame: Week 24
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 189 | 202 | 199
days | 1.3 (1.75) | 2.0 (2.24) | 1.8 (2.18)

44. Secondary Outcome: Amount of Rescue Medication Taken at Weeks 2, 4, 8, 12 and 16
Description: In case of inadequate pain relief , acetaminophen up to 3000 mg per day up to 3 days in a week could be taken as rescue medication. The total dosage of acetaminophen in milligrams used during the specified week were summarized.
Time Frame: Week 2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
milligrams
  Week 2 | 3226.0 (698.10) | 3139.1 (655.37) | 2537.6 (530.44)
  Week 4 | 3033.2 (774.34) | 2815.6 (703.90) | 2005.3 (484.54)
  Week 8 | 2608.6 (706.60) | 2385.9 (633.42) | 2104.2 (556.57)
  Week 12 | 2121.2 (698.93) | 1810.1 (567.14) | 1633.4 (506.13)
  Week 16 | 2303.7 (747.74) | 2846.9 (906.15) | 2166.0 (670.55)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 42, analysis 1]; Test type: Superiority; p = 0.9164, Negative binomial model; LS Mean Ratio = 0.97, 95% CI 2-sided [0.58 to 1.62], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5/5 mg; Test type: Superiority — [test comment as in outcome 42, analysis 2]; p = 0.3542, Negative binomial model; LS Mean Ratio = 0.79, 95% CI 2-sided [0.47 to 1.31], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 42, analysis 3]; Test type: Superiority; p = 0.8065, Negative binomial model; LS Mean Ratio = 0.93, 95% CI 2-sided [0.51 to 1.68], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 42, analysis 3]; Test type: Superiority; p = 0.1752, Negative binomial model; LS Mean Ratio = 0.66, 95% CI 2-sided [0.36 to 1.20], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 42, analysis 5]; Test type: Superiority; p = 0.7837, Negative binomial model; LS Mean Ratio = 0.91, 95% CI 2-sided [0.48 to 1.73], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 42, analysis 5]; Test type: Superiority; p = 0.5062, Negative binomial model; LS Mean Ratio = 0.81, 95% CI 2-sided [0.43 to 1.52], Standard Error of Mean 0.26
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 42, analysis 7]; Test type: Superiority; p = 0.6821, Negative binomial model; LS Mean Ratio = 0.85, 95% CI 2-sided [0.40 to 1.82], Standard Error of Mean 0.33
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 42, analysis 7]; Test type: Superiority; p = 0.5032, Negative binomial model; LS Mean Ratio = 0.77, 95% CI 2-sided [0.36 to 1.65], Standard Error of Mean 0.30
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 42, analysis 9]; Test type: Superiority; p = 0.5796, Negative binomial model; LS Mean Ratio = 1.24, 95% CI 2-sided [0.58 to 2.61], Standard Error of Mean 0.47
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5/5 mg; [analysis description as in outcome 42, analysis 9]; Test type: Superiority; p = 0.8725, Negative binomial model; LS Mean Ratio = 0.94, 95% CI 2-sided [0.44 to 2.00], Standard Error of Mean 0.36

45. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Week 40 that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to Week 40
Population: The safety population was defined as all participants treated with Tanezumab or placebo subcutaneously.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
Participants
  AEs | 145 | 156 | 143
  SAEs | 9 | 7 | 11

46. Secondary Outcome: Number of Participants With Treatment-Emergent Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Week 40 that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator.
Time Frame: Baseline up to Week 40
Population: The safety population was defined as all participants treated with Tanezumab or placebo subcutaneously.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
Participants
  AEs | 31 | 40 | 33
  SAEs | 0 | 0 | 0

47. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities With Regard to Normal Baseline
Description: Primary Abnormality criteria: hemoglobin; hematocrit; RBC count [less than{<}0.8* lower limit of normal[LLN]; Ery. mean corpuscular volume/ hemoglobin/ HGB concentration, erythrocytes distribution width <0.9*LLN, >1.1*ULN; platelets <0.5*LLN,>1.75*upper limit of normal (ULN); white blood cell count<0.6*LLN, >1.5*ULN; Lymphocytes,Leukocytes,Neutrophils <0.8*LLN, >1.2*ULN; Basophils, Eosinophils, Monocytes >1.2*ULN; Prothrombin time/Intl. normalized ratio >1.1*ULN; total bilirubin>1.5*ULN; aspartate aminotransferase, alanine aminotransferase, gamma GT,LDH, alkaline phosphatase >3.0*ULN; total protein; albumin<0.8*LLN, >1.2*ULN; blood urea nitrogen, creatinine, Cholesterol, triglycerides >1.3*ULN; Urate >1.2*ULN; sodium <0.95*LLN,>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate <0.9*LLN, >1.1*ULN; phosphate <0.8*LLN, >1.2*ULN; glucose <0.6*LLN, >1.5*ULN;Hemoglobin A1C >1.3*ULN; creatine kinase >2.0*ULN, specific gravity <1.003, >1.030; pH<4.5, >8; Urine Leukocytes >=20.
Time Frame: Baseline up to Week 40
Population: The safety population was defined as all participants treated with Tanezumab or placebo subcutaneously. Here "Overall number of participants analysed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 204 | 208 | 212
Participants | 20 | 12 | 11

48. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities With Regard to Abnormal Baseline
Description: Primary Abnormality criteria: hemoglobin; hematocrit; RBC count < 0.8*LLN; Ery. mean corpuscular volume/ hemoglobin/ HGB concentration, erythrocytes distribution width <0.9*LLN, >1.1*ULN; platelets <0.5*LLN,>1.75*upper limit of normal (ULN); white blood cell count<0.6*LLN, >1.5*ULN; Lymphocytes, Leukocytes, Neutrophils <0.8*LLN, >1.2*ULN; Basophils, Eosinophils, Monocytes >1.2*ULN; Prothrombin time/Intl. normalized ratio >1.1*ULN; total bilirubin>1.5*ULN; aspartate aminotransferase, alanine aminotransferase, gamma GT,LDH, alkaline phosphatase >3.0*ULN; total protein; albumin<0.8*LLN, >1.2*ULN; blood urea nitrogen, creatinine, Cholesterol, triglycerides >1.3*ULN; Urate >1.2*ULN; sodium <0.95*LLN,>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate <0.9*LLN, >1.1*ULN; phosphate <0.8*LLN, >1.2*ULN; glucose <0.6*LLN, >1.5*ULN; Hemoglobin A1C >1.3*ULN; creatine kinase >2.0*ULN; Urine erythrocytes >=20.
Time Frame: Baseline up to Week 40
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 161 | 158 | 166
Participants | 14 | 10 | 3

49. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at Weeks 2, 4, 8, 12, 16, 24, 40
Description: Measurement of BP included sitting systolic (SBP) and diastolic BP (DBP).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 40
Population: The safety population was defined as all participants treated with Tanezumab or placebo subcutaneously. Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
millimeters of mercury (mmHg)
  SBP: Baseline | 126.6 (11.11) | 126.4 (12.20) | 127.3 (12.85)
  SBP:Change at Week 2: number analyzed (Participants) | 224 | 226 | 227
  SBP:Change at Week 2 | -0.7 (10.77) | -1.8 (11.20) | -0.8 (11.12)
  SBP:Change at Week 4: number analyzed (Participants) | 222 | 227 | 226
  SBP:Change at Week 4 | -1.2 (10.98) | -2.2 (11.38) | -2.2 (11.89)
  SBP:Change at Week 8: number analyzed (Participants) | 207 | 221 | 221
  SBP:Change at Week 8 | -0.4 (12.12) | -1.7 (12.08) | -0.7 (12.06)
  SBP:Change at Week 12: number analyzed (Participants) | 199 | 217 | 210
  SBP:Change at Week 12 | -0.4 (13.90) | -3.8 (11.93) | -1.5 (12.33)
  SBP:Change at Week 16: number analyzed (Participants) | 189 | 207 | 208
  SBP:Change at Week 16 | -0.4 (10.79) | -1.8 (11.71) | -0.8 (12.52)
  SBP:Change at Week 24: number analyzed (Participants) | 182 | 196 | 201
  SBP:Change at Week 24 | 0.8 (12.05) | 0.1 (13.04) | 0.7 (11.89)
  SBP:Change at Week 40: number analyzed (Participants) | 179 | 191 | 190
  SBP:Change at Week 40 | 0.4 (12.61) | -0.9 (12.66) | -0.1 (11.30)
  DBP: Baseline | 77.7 (8.25) | 78.0 (8.47) | 77.9 (8.79)
  DBP:Change at Week 2: number analyzed (Participants) | 224 | 226 | 227
  DBP:Change at Week 2 | 0.2 (7.41) | -0.7 (7.60) | -0.6 (7.56)
  DBP:Change at Week 4: number analyzed (Participants) | 222 | 227 | 226
  DBP:Change at Week 4 | -0.7 (7.55) | -1.6 (8.36) | -1.3 (7.52)
  DBP:Change at Week 8: number analyzed (Participants) | 207 | 221 | 221
  DBP:Change at Week 8 | -0.4 (7.41) | -0.8 (7.90) | -0.1 (8.18)
  DBP:Change at Week 12: number analyzed (Participants) | 199 | 217 | 210
  DBP:Change at Week 12 | -0.3 (8.59) | -2.5 (8.13) | -1.2 (8.49)
  DBP:Change at Week 16: number analyzed (Participants) | 189 | 207 | 208
  DBP:Change at Week 16 | 0.2 (6.97) | -1.8 (7.97) | -1.0 (8.55)
  DBP:Change at Week 24: number analyzed (Participants) | 182 | 196 | 201
  DBP:Change at Week 24 | 0.5 (7.85) | -0.5 (8.74) | 0.2 (9.07)
  DBP:Change at Week 40: number analyzed (Participants) | 179 | 191 | 190
  DBP:Change at Week 40 | -1.4 (8.33) | -1.4 (9.64) | -0.6 (8.64)

50. Secondary Outcome: Change From Baseline in Heart Rate at Weeks 2, 4, 8, 12,16, 24, 40
Description: Heart rate was measured at sitting position.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24 and 40
Population: The safety population was defined as all participants treated with Tanezumab or placebo subcutaneously. Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified time points.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
beats per minute
  Baseline | 70.9 (8.96) | 71.4 (10.05) | 72.5 (9.76)
  Change at Week 2: number analyzed (Participants) | 224 | 226 | 227
  Change at Week 2 | 0.7 (7.71) | 1.1 (8.40) | 0.3 (8.12)
  Change at Week 4: number analyzed (Participants) | 222 | 227 | 226
  Change at Week 4 | 0.9 (7.76) | 0.5 (7.56) | 0.8 (8.60)
  Change at Week 8: number analyzed (Participants) | 207 | 221 | 221
  Change at Week 8 | 0.2 (8.65) | -0.3 (8.33) | -0.1 (7.91)
  Change at Week 12: number analyzed (Participants) | 199 | 217 | 210
  Change at Week 12 | 0.6 (8.24) | 1.1 (8.07) | 0.0 (8.81)
  Change at Week 16: number analyzed (Participants) | 189 | 207 | 208
  Change at Week 16 | -0.0 (8.47) | 0.3 (8.82) | -0.6 (8.32)
  Change at Week 24: number analyzed (Participants) | 182 | 196 | 201
  Change at Week 24 | 0.7 (9.11) | 0.4 (8.56) | 0.6 (8.42)
  Change at Week 40: number analyzed (Participants) | 179 | 191 | 190
  Change at Week 40 | 0.7 (8.72) | 0.5 (10.11) | 0.2 (8.49)

51. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters at Weeks 16 and 40
Description: A 12-lead ECG was recorded after participants had rested for at least 5 minutes in the supine position in a quiet environment. All standard intervals (PR, QRS, QT, QTcF, QTcB, QTcF, RR intervals) were collected.
Time Frame: Baseline, Weeks 16, 40
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
millisecond
  RR Interval: Baseline: number analyzed (Participants) | 232 | 231 | 232
  RR Interval: Baseline | 932.4 (137.58) | 927.3 (140.92) | 911.0 (128.93)
  RR Interval:Change at Week 16: number analyzed (Participants) | 187 | 204 | 206
  RR Interval:Change at Week 16 | -20.4 (114.08) | -13.1 (119.83) | -10.1 (115.78)
  RR Interval:Change at Week 40: number analyzed (Participants) | 179 | 191 | 188
  RR Interval:Change at Week 40 | -31.6 (113.49) | -28.5 (116.77) | -22.1 (114.23)
  PR Interval: Baseline: number analyzed (Participants) | 226 | 229 | 231
  PR Interval: Baseline | 168.4 (26.20) | 163.2 (25.73) | 162.9 (26.83)
  PR Interval:Change at Week 16: number analyzed (Participants) | 183 | 202 | 204
  PR Interval:Change at Week 16 | -1.7 (12.17) | 1.8 (12.08) | -0.3 (12.41)
  PR Interval:Change at Week 40: number analyzed (Participants) | 176 | 189 | 186
  PR Interval:Change at Week 40 | -0.9 (13.63) | -1.2 (13.37) | -0.3 (12.65)
  QRS Interval: Baseline: number analyzed (Participants) | 232 | 231 | 232
  QRS Interval: Baseline | 94.8 (14.63) | 94.6 (11.69) | 93.8 (12.56)
  QRS Interval:Change at Week 16: number analyzed (Participants) | 187 | 204 | 206
  QRS Interval:Change at Week 16 | -0.3 (6.53) | -0.4 (7.47) | -1.1 (6.99)
  QRS Interval:Change at Week 40: number analyzed (Participants) | 179 | 191 | 188
  QRS Interval:Change at Week 40 | -0.9 (7.36) | -0.7 (7.71) | -1.6 (7.76)
  QT Interval: Baseline: number analyzed (Participants) | 232 | 191 | 232
  QT Interval: Baseline | 401.3 (27.20) | 401.5 (28.82) | 397.9 (26.26)
  QT Interval:Change at Week 16: number analyzed (Participants) | 186 | 204 | 206
  QT Interval:Change at Week 16 | -2.7 (21.24) | -1.7 (22.08) | -1.8 (21.20)
  QT Interval:Change at Week 40: number analyzed (Participants) | 179 | 191 | 188
  QT Interval:Change at Week 40 | -6.1 (21.14) | -6.1 (20.67) | -6.3 (22.68)
  QTCB Interval: Baseline: number analyzed (Participants) | 232 | 231 | 232
  QTCB Interval: Baseline | 417.4 (21.67) | 418.8 (20.45) | 418.7 (21.55)
  QTCB Interval:Change at Week 16: number analyzed (Participants) | 186 | 204 | 206
  QTCB Interval:Change at Week 16 | 1.9 (16.59) | 1.2 (17.25) | 0.4 (17.52)
  QTCB Interval:Change at Week 40: number analyzed (Participants) | 179 | 191 | 188
  QTCB Interval:Change at Week 40 | 1.1 (15.97) | 0.3 (17.60) | -2.0 (16.43)
  QTCF Interval: Baseline: number analyzed (Participants) | 232 | 231 | 232
  QTCF Interval: Baseline | 411.8 (18.93) | 412.7 (18.36) | 411.4 (18.84)
  QTCF Interval:Change at Week 16: number analyzed (Participants) | 186 | 204 | 206
  QTCF Interval:Change at Week 16 | 0.3 (13.85) | 0.2 (14.54) | -0.4 (14.44)
  QTCF Interval:Change at Week 40: number analyzed (Participants) | 179 | 191 | 188
  QTCF Interval:Change at Week 40 | -1.4 (13.40) | -1.9 (14.08) | -3.5 (14.34)

52. Secondary Outcome: Change From Baseline in Heart Rate (as Assessed by ECG) at Weeks 16 and 40
Time Frame: Baseline, Weeks 16 and 40
Population: The safety population was defined as all participants treated with Tanezumab or placebo subcutaneously. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
beats per minute
  Baseline: number analyzed (Participants) | 232 | 231 | 232
  Baseline | 65.8 (9.78) | 66.3 (10.97) | 67.2 (9.80)
  Change at Week 16: number analyzed (Participants) | 187 | 204 | 206
  Change at Week 16 | 1.3 (8.68) | 0.9 (8.81) | 0.8 (8.74)
  Change at Week 40: number analyzed (Participants) | 179 | 191 | 188
  Change at Week 40 | 2.5 (8.55) | 2.2 (9.13) | 1.5 (8.88)

53. Secondary Outcome: Percentage of Participants With Adjudicated Joint Safety Outcomes
Description: Incidence of participants with any of the joint safety adjudication outcomes of primary osteonecrosis, rapidly progressive osteoarthritis (OA) (type 1 and type 2), subchondral insufficiency fracture (or SPONK), or pathological fracture.
Time Frame: Baseline up to Week 40
Population: The safety population was defined as all participants treated with Tanezumab or placebo subcutaneously. Here, 'Overall number of participants analyzed' signifies participants analyzed by adjudication committee.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 5 | 14 | 18
percentage of participants
  Composite Joint Safety Endpoint | 0 [0.0 to 1.6] | 2.2 [0.7 to 5.0] | 0.4 [0.0 to 2.4]
  Rapidly Progressive OA | 0 [0.0 to 1.6] | 2.2 [0.7 to 5.0] | 0.4 [0.0 to 2.4]
  Rapidly Progressive OA type 1 | 0 [0.0 to 1.6] | 1.3 [0.3 to 3.7] | 0.4 [0.0 to 2.4]
  Rapidly Progressive OA type 2 | 0 [0.0 to 1.6] | 0.9 [0.1 to 3.1] | 0.0 [0.0 to 1.6]
  Primary Osteonecrosis | 0 [0.0 to 1.6] | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Pathological Fracture | 0 [0.0 to 1.6] | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]
  Subchondral Insufficiency Fracture | 0 [0.0 to 1.6] | 0 [0.0 to 1.6] | 0 [0.0 to 1.6]

54. Secondary Outcome: Percentage of Participants With Total Joint Replacements
Description: Percentage of participants who underwent total knee, hip or shoulder joint replacement surgery.
Time Frame: Baseline up to Week 40
Population: The safety population was defined as all participants treated with Tanezumab or placebo subcutaneously.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
percentage of participants | 1.7 [0.5 to 4.4] | 3.5 [1.5 to 6.7] | 6.9 [4.0 to 10.9]

55. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 8,12,16, 24 and 40
Description: NIS is a standardized instrument used to evaluate participant for signs of peripheral neuropathy. NIS is the sum of scores of 37 items, from both the left and right side, where 24 items scored from 0 (normal) to 4 (paralysis), higher score indicated higher abnormality/impairment and 13 items scored from 0 (normal), 1 (decreased) and 2 (absent), higher score indicated higher impairment. NIS possible overall score ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicated increased impairment.
Time Frame: Baseline, Weeks 2, 4, 8,12,16, 24 and 40
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Baseline | 1.09 (2.60) | 2.01 (4.75) | 1.80 (4.50)
  Change at Week 2: number analyzed (Participants) | 221 | 224 | 224
  Change at Week 2 | -0.21 (1.38) | -0.14 (1.64) | -0.31 (1.59)
  Change at Week 4: number analyzed (Participants) | 227 | 229 | 228
  Change at Week 4 | -0.17 (1.50) | -0.15 (2.37) | -0.32 (1.88)
  Change at Week 8: number analyzed (Participants) | 229 | 230 | 229
  Change at Week 8 | -0.14 (1.55) | -0.22 (2.06) | -0.16 (1.73)
  Change at Week 12: number analyzed (Participants) | 229 | 230 | 229
  Change at Week 12 | -0.14 (1.70) | -0.31 (2.37) | -0.28 (2.24)
  Change at Week 16: number analyzed (Participants) | 229 | 230 | 229
  Change at Week 16 | -0.20 (1.71) | -0.24 (2.28) | -0.35 (2.72)
  Change at Week 24: number analyzed (Participants) | 229 | 230 | 229
  Change at Week 24 | -0.27 (1.73) | -0.16 (1.83) | -0.29 (2.60)
  Change at Week 40: number analyzed (Participants) | 229 | 230 | 229
  Change at Week 40 | -0.25 (1.71) | -0.25 (2.16) | -0.52 (2.55)

56. Secondary Outcome: Number of Participants With Confirmed Orthostatic Hypotension
Description: Orthostatic hypotension was defined as postural change (supine to standing) that met the following criteria: For systolic BP <=150 mmHg (mean supine): Reduction in systolic BP>=20 mmHg or reduction in diastolic BP>=10 mmHg at the 1 and/or 3 minute standing BP measurements. For systolic BP >150 mmHg (mean supine): Reduction in systolic BP>=30 mmHg or reduction in diastolic BP>=15 mmHg at the 1 and/or 3 minute standing BP measurements. If the 1 minute or 3 minute standing BP in a sequence met the orthostatic hypotension criteria, then that sequence was considered positive. If 2 of 2 or 2 of 3 sequences were positive, then orthostatic hypotension was considered confirmed.
Time Frame: Baseline up to Week 40
Population: The safety population was defined as all participants treated with Tanezumab or placebo subcutaneously. Here, 'Overall number of participants analyzed' signifies participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 227 | 230 | 228
Participants | 1 | 3 | 1

57. Secondary Outcome: Change From Baseline in Survey of Autonomic Symptom (SAS) Scores at Weeks 24 and 40
Description: The SAS is a 12 item (11 for females) questionnaire, from which the total number of symptoms (0-12 for males and 0-11 for females) is calculated. Each positive symptom is rated from 1 (not at all) to 5 (a lot). The total impact score was the sum of all symptom rating scores, with 0 assigned where the participant did not have the particular symptom. The range for the total impact score is 0-60 for males and 0-55 for females, higher scores indicating higher impact.
Time Frame: Baseline, Weeks 24 and 40
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
units on a scale
  Number of symptoms reported: Baseline | 0.47 (0.71) | 0.54 (0.82) | 0.45 (0.73)
  Number of symptoms reported: Change at Week 24: number analyzed (Participants) | 182 | 197 | 201
  Number of symptoms reported: Change at Week 24 | 0.42 (1.33) | 0.30 (1.25) | 0.38 (1.26)
  Number of symptoms reported: Change at Week 40: number analyzed (Participants) | 178 | 190 | 191
  Number of symptoms reported: Change at Week 40 | 0.23 (1.22) | 0.18 (1.27) | 0.26 (1.28)
  Total Symptom Impact Score: Baseline | 1.07 (1.72) | 1.15 (1.71) | 1.00 (1.73)
  Total Symptom Impact Score: Change at Week 24: number analyzed (Participants) | 182 | 197 | 201
  Total Symptom Impact Score: Change at Week 24 | 1.44 (3.82) | 1.22 (3.66) | 1.22 (3.48)
  Total Symptom Impact Score: Change at Week 40: number analyzed (Participants) | 178 | 190 | 191
  Total Symptom Impact Score: Change at Week 40 | 0.83 (3.43) | 0.89 (3.79) | 0.96 (3.46)

58. Secondary Outcome: Number of Participants With Anti-Tanezumab Antibodies
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using a semi quantitative enzyme linked immunosorbent assay (ELISA). Participants listed as having anti-tanezumab antibodies had ADA titer level >=3.32. Less than 3.32 was considered below the limit of quantitation.
Time Frame: Baseline, Weeks 8,16, 24 and 40
Population: as for outcome 52
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
Number analyzed (Participants) | 232 | 231 | 233
Participants
  Baseline: number analyzed (Participants) | 230 | 227 | 229
  Baseline | 25 | 25 | 23
  Week 8: number analyzed (Participants) | 206 | 217 | 217
  Week 8 | 22 | 29 | 36
  Week 16: number analyzed (Participants) | 189 | 206 | 204
  Week 16 | 16 | 35 | 43
  Week 24: number analyzed (Participants) | 182 | 193 | 199
  Week 24 | 15 | 30 | 40
  Week 40: number analyzed (Participants) | 178 | 189 | 187
  Week 40 | 18 | 29 | 33

ADVERSE EVENTS:
Time Frame: Baseline up to Week 40 (end of study)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as nonserious in another participant or 1 participant may have experienced both serious and nonserious event during study.
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 2.5/5 mg
All-Cause Mortality (participants affected / at risk) | 0/232 | 0/231 | 2/233
Serious Adverse Events (participants affected / at risk) | 9/232 | 7/231 | 11/233
Other Adverse Events (participants affected / at risk) | 143/232 | 155/231 | 141/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=232) | Tanezumab 2.5 mg (N=231) | Tanezumab 2.5/5 mg (N=233)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 2
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Abdominal hernia infection (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Prostatectomy (Surgical and medical procedures) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=232) | Tanezumab 2.5 mg (N=231) | Tanezumab 2.5/5 mg (N=233)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 3 | 3 | 2
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 4 | 1 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 2 | 3 | 0
Dry eye (Eye disorders) | 0 | 3 | 2
Eye pruritus (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 3
Defaecation urgency (Gastrointestinal disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 3 | 0 | 2
Dental paraesthesia (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 3 | 1 | 1
Feeling hot (General disorders) | 0 | 2 | 0
Injection site erythema (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 1 | 1
Injection site reaction (General disorders) | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 5 | 7
Pain (General disorders) | 1 | 0 | 2
Peripheral swelling (General disorders) | 2 | 0 | 3
Pyrexia (General disorders) | 2 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 5 | 1 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 3 | 1
Peripheral coldness (Vascular disorders) | 0 | 1 | 3
Dental prosthesis placement (Surgical and medical procedures) | 1 | 0 | 0
Foot operation (Surgical and medical procedures) | 0 | 0 | 1
Gingival graft (Surgical and medical procedures) | 0 | 0 | 1
Nail operation (Surgical and medical procedures) | 0 | 0 | 1
Toe operation (Surgical and medical procedures) | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 2
Tooth repair (Surgical and medical procedures) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Acarodermatitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 5 | 8 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 3 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 1
Diarrhoea infectious (Infections and infestations) | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2
Epicondylitis (Injury, poisoning and procedural complications) | 2 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 2
Blood urea increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 2 | 0 | 0
International normalised ratio decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 1 | 1
White blood cell count increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 4 | 2 | 3
Anxiety (Psychiatric disorders) | 2 | 0 | 1
Depression (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 3
Irritability (Psychiatric disorders) | 0 | 0 | 1
Sleep disorder due to general medical condition, insomnia type (Psychiatric disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Decreased vibratory sense (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 3 | 4
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 10 | 9 | 9
Hypoaesthesia (Nervous system disorders) | 6 | 5 | 6
Migraine (Nervous system disorders) | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 8 | 3
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 3 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Gingival abscess (Infections and infestations) | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 4 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 5 | 5 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 16 | 20 | 17
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 2 | 1 | 1
Postoperative wound infection (Infections and infestations) | 2 | 1 | 0
Sinobronchitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 5 | 6 | 3
Skin infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 2 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 11 | 10
Urinary tract infection (Infections and infestations) | 2 | 4 | 4
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 1
Wound infection bacterial (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 13 | 10
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 3 | 2
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 5 | 4
Limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 5 | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 5 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 4 | 4
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Repetitive strain injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 34 | 34
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 13 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint noise (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 5 | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 | 9 | 6
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 17 | 8
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 9 | 9
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 2
Acid peptic disease (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 1
Thirst (General disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Artificial crown procedure (Surgical and medical procedures) | 1 | 0 | 0
Blepharoplasty (Surgical and medical procedures) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Wound abscess (Infections and infestations) | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Subchondral insufficiency fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Skin neoplasm excision (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 1
Viral rhinitis (Infections and infestations) | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Breast haematoma (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 1 | 0
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT02697773/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT02697773/SAP_001.pdf